Objective Vision Evaluation of Two Cosmetic Contact Lenses

Protocol CR-6396

Version: 2.0

Date: 29 January 2020

Investigational Products: etafilcon A with PVP cosmetic lenses, 1-DAY ACUVUE® DEFINE® Radiant Sweet<sup>TM</sup> contact Lenses

Key Words: etafilcon A with PVP cosmetic lenses, 1-DAY ACUVUE® DEFINE® Radiant Sweet<sup>TM</sup>, daily disposable, logMAR visual acuity, objective vision

#### Statement of Compliance to protocol, GCP and applicable regulatory guidelines:

This trial will be conducted in compliance with the protocol, ISO 14155,<sup>1</sup> the International Conference on Harmonization Good Clinical Practice E6 (ICH-GCP),<sup>2</sup> the Declaration of Helsinki,<sup>3</sup> and all applicable regulatory requirements.

#### **Confidentiality Statement:**

This document contains confidential information, which should not be copied, referred to, released or published without written approval from Johnson & Johnson Vision Care, Inc. The information may not be disclosed to others except to the extent necessary to obtain Institutional Review Board/Independent Ethics Committee approval and informed consent, or as required by International, Federal and State Laws, as applicable. Persons to whom this information is disclosed must be informed that this information is privileged and confidential and that it should not be further disclosed without the written permission of Johnson & Johnson Vision Care, Inc. Any supplemental information that may be added to this document is also confidential and proprietary to Johnson & Johnson Vision Care, Inc. and must be kept in confidence in the same manner as the contents of this document.

| TABL | E OF CONTENTS | |
|---|---|---|
| PROTO | DCOL TITLE, NUMBER, VERSION | 6 |
| SPONS | SOR NAME AND ADDRESS | 6 |
| MEDIC | CAL MONITOR | 6 |
| AUTH | ORIZED SIGNATURES | 7 |
| CHAN | GE HISTORY | 8 |
| SYNO | PSIS | 9 |
| COMM | MONLY USED ABBREVIATIONS AND DEFINITIONS OF TERMS | 14 |
| 1. IN | TRODUCTION AND BACKGROUND | 15 |
| 1.1. | Name and Descriptions of Investigational Products | 15 |
| 1.2. | Intended Use of Investigational Products | 15 |
| 1.3. | Summary of Findings from Nonclinical Studies | 15 |
| 1.4. | Summary of Known Risks and Benefits to Human Subjects | 16 |
| 1.5.<br>Stud | | d Clinical |
| 2. ST | TUDY OBJECTIVES, ENDPOINTS AND HYPOTHESES | 17 |
| 2.1. | Objectives | 17 |
| 2.2. | Endpoints | 17 |
| 2.3. | Hypotheses | 19 |
| 3. TA | ARGETED STUDY POPULATION | 19 |
| 3.1. | General Characteristics | 19 |
| 3.2. | Inclusion Criteria. | 19 |
| 3.3. | Exclusion Criteria. | 20 |
| 3.4. | Enrollment Strategy | 20 |
| 4. ST | TUDY DESIGN AND RATIONALE | 20 |
| 4.1. | Description of Study Design | 20 |
| 4.2. | Study Design Rationale | 21 |
| 4.3. | Enrollment Target and Study Duration | 21 |
| 5. TI | EST ARTICLE ALLOCATION AND MASKING | 21 |
| 5.1. | Test Article Allocation | 21 |
| 5.2. | Masking | 21 |
| 5.3. | Procedures for Maintaining and Breaking the Masking | 22 |
| 6. ST | TUDY INTERVENTION | 22 |
| 6.1 | Identity of Test Articles | 22 |

| 6.2 | 2. A | Ancillary Supplies/Products | 23 |
|---|---|---|---|
| 6.3 | 8. A | Administration of Test Articles | 24 |
| 6.4 | l. P | ackaging and Labeling | 24 |
| 6.5 | 5. S | torage Conditions | 24 |
| 6.6 | 5. C | Collection and Storage of Samples | 24 |
| 6.7 | . A | Accountability of Test Articles | 24 |
| 7. | STUI | DY EVALUATIONS | 25 |
| 7.1 | . Т | ime and Event Schedule | 25 |
| 7.2 | 2. E | Detailed Study Procedures | 26 |
| VISI | Г1 | | 26 |
| | FINA | L EVALUATION | 37 |
| 7.3 | . t | Jnscheduled Visits | 38 |
| 7.4 | l. L | aboratory Procedures | 39 |
| 8. | SUB. | JECTS COMPLETION/WITHDRAWAL | 39 |
| 8.1 | . ( | Completion Criteria | 39 |
| 8.2 | 2. V | Vithdrawal/Discontinuation from the Study | 39 |
| 9. | PRE- | STUDY AND CONCOMITANT INTERVENTION/MEDICATION | 40 |
| 9.1 | . S | ystemic Medications | 40 |
| 10. | DE | VIATIONS FROM THE PROTOCOL | 40 |
| 11. | STU | UDY TERMINATION | 41 |
| 12. | PR | OCEDURE FOR HANDLING PRODUCT QUALITY COMPLAINTS | 41 |
| 13. | AD | VERSE EVENTS | 43 |
| 13. | .1. | Definitions and Classifications | 43 |
| 13. | .2. | Assessing Adverse Events | 45 |
| 13. | 2.1. | Causality Assessment | 45 |
| 13. | .2.2. | Severity Assessment | 45 |
| 13. | .3. | Documentation and Follow-Up of Adverse Events | 46 |
| 13. | .4. | Reporting Adverse Events | 47 |
| 13. | .4.1. | Reporting Adverse Events to Sponsor | 47 |
| 13. | .4.2. | Reporting Adverse Events to the Responsible IEC/IRB and Health Authorities . | 48 |
| 13. | .4.3. | Event of Special Interest | 48 |
| 13. | .5. | Reporting of Pregnancy | 48 |
| 14. | STA | ATISTICAL METHODS | 49 |
| 14. | .1. | General Considerations | 49 |

| 14.2. | Sample Size Justification | 49 |
|---|---|---|
| 14.3. | Analysis Populations | 49 |
| 14.4. | Level of Statistical Significance | 49 |
| 14.5. | Primary Analysis | 49 |
| 14.6. | Secondary Analysis | 50 |
| 14.7. | Other Exploratory Analyses | 50 |
| 14.8. | Interim Analysis | 50 |
| 14.9. | Procedure for Handling Missing Data and Drop-Outs | 50 |
| 14.10. | Procedure for Reporting Deviations from Statistical Plan | 50 |
| 15. DA | TA HANDLING AND RECORD KEEPING/ARCHIVING | 50 |
| 15.1. | Electronic Case Report Form/Data Collection | 50 |
| 15.2. | Subject Record | 51 |
| 15.3 | ClinicalTrials.gov | 51 |
| 16. DA | TA MANAGEMENT | 51 |
| 16.1. | Access to Source Data/Document | 51 |
| 16.2. | Confidentiality of Information. | 51 |
| 16.3. | Data Quality Assurance | 52 |
| 17. CL | INICAL MONITORING | 52 |
| 18. ET. | HICAL AND REGULATORY ASPECTS | 53 |
| 18.1. | Study-Specific Design Considerations | 53 |
| 18.2. | Investigator Responsibility | 53 |
| 18.3. | Independent Ethics Committee or Institutional Review Board (IEC/IRB) | 53 |
| 18.4. | Informed Consent | 54 |
| 18.5. | Privacy of Personal Data | 55 |
| 19. ST | UDY RECORD RETENTION | 56 |
| 20. FIN | VANCIAL CONSIDERATIONS | 57 |
| 21. PU | BLICATION | 57 |
| 22. RE | FERENCES | 58 |
| APPEND | IX A: PATIENT REPORTED OUTCOMES (STUDY QUESTIONNAIRES) | 59 |
| APPEND | IX B: PATIENT INSTRUCTION GUIDE | 64 |
| APPEND | IX C: PACKAGE INSERT (APPROVED PRODUCT) | 65 |
| APPEND | | |
| | Near LogMAR Visual Acuity Measurement Procedure | 69 |
| | Lens Fitting Characteristics | 72 |

| Subject Reported Ocular Symptoms/Problems | 79 |
|--------------------------------------------------------------------|-----|
| Determination of Distance Spherocylindrical Refractions | 81 |
| Biomicroscopy Scale | 88 |
| , Distance and Near Visual Acuity Evaluation | |
| Distance LogMAR Visual Acuity Measurement Procedure | |
| Measuring Pupil Diameter with NeurOptics VIP-200 Variable Pupillom | |
| Visual Acuity Chart Luminance and Room Illumination Testing | 107 |
| Qcsf Contrast Sensitivity | 113 |
| APPENDIX E: WORK AID: AST qVA-Custom 100 | |
| APPENDIX F: WAVEFRONT AND TOPOGRAPHY MEASUREMENT USING V<br>VX118 | |
| APPENDIX G: COSMETIC FIT AND HULA HOOP | |
| APPENDIX H: VISUAL EXPERIENCE WORK AID | 144 |
| PROTOCOL COMPLIANCE INVESTIGATOR(S) SIGNATURE PAGE | |
| TABLE OF CONTENTS Figure 1: Study Flowchart | 13 |
| TABLE OF CONTENTS | |
| Table 1: Test Articles | |
| Table 2: Ancillary Supplies | |
| 1 auto 3. 1 mio ana 12 vento | 43 |

#### PROTOCOL TITLE, NUMBER, VERSION

Title: Objective Vision Evaluation of Two Cosmetic Contact Lenses

Protocol Number: CR-6396

Version: 2.0

Date: 29 January 2020

#### SPONSOR NAME AND ADDRESS

Johnson & Johnson Vision Care (JJVC) 7500 Centurion Parkway Jacksonville, FL 32256

#### MEDICAL MONITOR

Name: Meredith Bishop OD, MS, FAAO Title: Senior Principal Research Optometrist Address: 7500 Centurion Parkway, Suite 100

Email: mbishop4@its.jnj.com

The Medical Monitor must be notified by the clinical institution/site by e-mail, fax, or telephone within 24 hours of learning of a Serious Adverse Event. The Medical Monitor may be contacted during business hours for adverse event questions. General study related questions should be directed towards your assigned clinical research associate.

The Medical Monitoring Plan is maintained as a separate document and included in the Trial Master File.

#### AUTHORIZED SIGNATURES

The signatures below constitutes the approval of this protocol and the attachments and provide the necessary assurances that this trial will be conducted according to all stipulations of the protocol, including all statements regarding confidentiality, and according to local legal and regulatory requirements and applicable U.S. federal regulations, ICH guidelines, ISO 14155, and the Declaration of Helsinki.

| Author/Study | | |
|---------------------|----------------------------------------|-------|
| Responsible | | |
| Clinician | See Electronic Signature Report | |
| | Meredith Bishop, OD, MS, FAAO | DATE |
| | Senior Principal Research Optometrist, | |
| | Clinical Science, R&D | |
| | , | |
| Clinical Operations | | |
| Manager | See Electronic Signature Report | |
| | 1 | DATE |
| | - | Dill |
| | Clinical Operations, R&D | |
| | cimical operations, recep | |
| Biostatistician | See Electronic Signature Report | |
| | I | DATE |
| | | DITTE |
| | Clinical Science, R&D | |
| | , | |
| Data Management | See Electronic Signature Report | |
| | ī | DATE |
| | Data and Systems, R&D | |
| Reviewer | See Electronic Signature Report | P 92 |
| | | DATE |
| | Research Fellow | |
| Approver | See Electronic Signature Report | |
| | | DATE |
| | Director, Specialty Growth | |
| | R&D | |

### **CHANGE HISTORY**

| Version | Originator | Description of Change(s) and Section<br>Number(s) Affected | Date |
|---|---|---|---|
| 1.0 | Meredith Bishop | Original Protocol | 24 January<br>2020 |
| 2.0 | Meredith Bishop | Updated Appendix E to include Work<br>Aid: AST qVA-Custom 100 | 29 January<br>2020 |

### **SYNOPSIS**

| Protocol Title | Objective Vision Evaluation of Two Cosmetic Contact |
|---|---|
| | Lenses |
| Sponsor | JJVC, 7500 Centurion Parkway, Jacksonville, FL 32256 |
| Clinical Phase | Confirmatory, Phase 3 |
| Trial Registration | This study will be registered on ClinicalTrials.gov based on |
| | the following: confirmatory study meets the requirements for |
| | registration. |
| Test Article(s) | Investigational Products: etafilcon A with cosmetic pattern |
| 2.5 | Approved Products: 1-DAY ACUVUE® DEFINE® Radiant |
| | Sweet <sup>TM</sup> |
| Wear and Replacement | Wear Schedule: Daily Wear |
| Schedules | Replacement Schedule: Daily Disposable |
| Objectives | Primary Objective |
| , | The primary objective of this study is to assess the objective |
| | vision of the study lenses at fitting. |
| | , |
| | Exploratory Objective |
| | Additional objectives include assessments of wavefront |
| | aberrometry, pupillometry, lens fit, subject reported ocular |
| | symptoms, and slit-lamp findings |
| Study Endpoints | Primary endpoints: |
| Study Emaponics | Distance logMAR visual acuity using ETDRS charts |
| | I Distance registrate visital desiry asing 2121ts character |
| | 2. Near logMAR visual acuity |
| | 3. qCSF |
| | 4. qVA |
| | 4. qvA |
| | Other observations will include: |
| | 1. Subjective Comfort, Vision via the CLUE <sup>5</sup> |
| | questionnaire |
| | 2. Visionix wavefront aberrometry |
| | 3. Pupillometry |
| | 4. Mechanical Lens fit |
| | 5. Cosmetic Lens fit/Hula Hoop |
| | 6. Ocular Physiology |
| Study Design | This is a single visit, single site, brand-masked, non- |
| , | dispensing, 2×2 bilateral crossover study. Each subject will |
| | be bilaterally fitted with one of the two test articles in each of |
| | the study periods. |
| | See the flow chart at the end of the synopsis table for the |
| | schematic of the study visits and procedures of main |
| | observations. |

| Sample Size | Up to 30 subjects will be enrolled with the aim of |
|---|---|
| | approximately 25 subjects completing. |
| Study Duration | The study is expected to last up to 1 month. The enrollment |
| | period will also be up to 2 weeks. |
| Anticipated Study | We will aim to recruit up to 30 habitual contact lens wearing |
| Population | subjects, ages 18 to 39 (inclusive). We will aim to enroll |
| 1 1 1 2 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 | female subjects ages 18-29. |
| Eligibility Criteria | |
| | Potential subjects must satisfy all of the following criteria to be enrolled in the study: 1. The subject must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form 2. Appear able and willing to adhere to the instructions set forth in this clinical protocol 3. Subjects between 18 and 39 (inclusive) years of age at the time of screening 4. Be a current soft contact lens wearer in both eyes with a minimum of 6 hours/day and 5 days/week over the last month by self-report 5. The subject must be willing to be photographed and/or video-taped Eligibility after Baseline: 6. The subject's vertex corrected spherical equivalent distance refraction must be in the range of -1.00 D to -5.00 D (inclusive) in each eye 7. The subject's refractive cylinder must be less than or equal to 0.75 D (inclusive) in each eye 8. Have spherical best corrected visual acuity of 20/25 or better in each eye |

| | I D |
|---|---|
| | Potential subjects who meet any of the following criteria will |
| | be excluded from participating in the study: |
| | 1. Currently pregnant or lactating |
| | 2. Any systemic disease (eg, Sjögren's Syndrome), allergies, infectious disease (eg, hepatitis, |
| | allergies, infectious disease (eg, hepatitis, tuberculosis), contagious immunosuppressive diseases |
| | (eg, HIV), autoimmune disease (eg rheumatoid |
| | arthritis), or other diseases, by self-report, which are |
| | known to interfere with contact lens wear and/or |
| | participation in the study (at the investigators |
| | discretion) |
| | 3. Use of systemic medications (eg, chronic steroid use) |
| | that are known to interfere with contact lens wear (at the investigators discretion) |
| | 4. Any previous, or planned (during the study) ocular |
| | surgery (eg, radial keratotomy, PRK, LASIK, etc.) |
| | 5. Participation in any contact lens or lens care product |
| | clinical trial within seven (7) days prior to study |
| | enrollment. |
| | 6. Employee or family members of clinical site (eg, |
| | Investigator, Coordinator, Technician) Exclusion |
| | Criteria after Baseline |
| | Eligibility after Baseline: |
| | 7. Any ocular allergies, infections or other ocular |
| | abnormalities that are known to interfere with contact |
| | lens wear and/or participation in the study. This may |
| | include, but not be limited to entropion, ectropion, |
| | extrusions, chalazia, recurrent styes, glaucoma, history |
| | of recurrent corneal erosions, aphakia, or corneal distortion (at the investigators discretion) |
| | 8. Clinically significant (Grade 3 or 4 on FDA scale) |
| | tarsal abnormalities, bulbar injection, corneal edema, |
| | corneal vascularization, corneal staining, or any other |
| | abnormalities of the cornea which would |
| | contraindicate contact lens wear. |
| Disallowed | None |
| Medications/Interventions | |
| Measurements and | logMAR visual acuity, qVA, qCSF, wavefront aberrometry, |
| Procedures | PRO questionnaires (comfort, vision, and handling), lens fit |
| | assessment, cosmetic lens fit assessment/hula hoop |
| | assessment, and safety parameters (slit lamp findings, |
| Microbiology or Other | entrance/exit visual acuity). None |
| Laboratory Testing | Tione |
| Laboratory resuing | |

| Study Termination | The occurrence of one or more Unanticipated Adverse |
|---|---|
| | Device Effect (UADE), or any SAE where relationship to |
| | study agent cannot be ruled out, will result in stopping |
| | further dispensing investigational product. In the event of a |
| | UADE or SAE, the Sponsor Medical Monitor may unmask |
| | the treatment regimen of subject(s) and may discuss this with |
| | the Principal Investigator before any further subjects are |
| | enrolled. |
| Ancillary Supplies/ Study- | Tears Naturale re-wetting drops, FluStrips fluorescein strips, |
| Specific Materials | Bausch & Lomb Sensitive Eyes plus Saline, or alternative |
| Section 1. The section of the sectio | products approved by the Sponsor. |
| Principal Investigator(s) | A full list of Principal Investigators, clinical sites, and |
| and Study | institutions is kept separately from the Study Protocol and is |
| Institution(s)/Site(s) | included in the study Trial Master File. |

Figure 1: Study Flowchart



^only with lens #1

#### COMMONLY USED ABBREVIATIONS AND DEFINITIONS OF TERMS

ADD Plus Power Required For Near Use

ADE Adverse Device Effect

AE Adverse Event/Adverse Experience
BCVA Best Corrected Visual Acuity

BSCVA Best Spectacle Corrected Visual Acuity

CFR Code of Federal Regulations
CLUE Contact Lens User Experience

COAS Complete Ophthalmic Analysis System

COM Clinical Operations Manager CRA Clinical Research Associate

CRF Case Report Form

CRO Contract Research Organization

CT Center Thickness

D Diopter

DMC Data Monitoring Committee eCRF Electronic Case Report Form EDC Electronic Data Capture

ETDRS Early Treatment Diabetic Retinopathy Study

FDA Food and Drug Administration

GCP Good Clinical Practice

HIPAA Health Insurance Portability and Accountability Act

IB Investigator's Brochure ICF Informed Consent Form

ICH International Conference on Harmonization

IDE Investigational Device Exemption
IEC Independent Ethics Committee
IRB Institutional Review Board

ISO International Organization for Standardization

ITT Intent-to-Treat

JJVC Johnson & Johnson Vision Care, Inc.

LC Limbus Center

LogMAR Logarithm of Minimal Angle of Resolution
MedDRA® Medical Dictionary for Regulatory Activities

MOP Manual of Procedures

NIH National Institutes of Health

OD Right Eye

OHRP Office for Human Research Protections
OHSR Office for Human Subjects Research

OS Left Eye
OU Both Eyes

PD Protocol Deviation

PHI Protected Health Information

PI Principal Investigator

PIG Patient Instruction Guide PQC Product Quality Complaint PRO Patient Reported Outcome

QA Quality Assurance QC Quality Control

qCSF Quick Contrast Sensitivity Function

qVA Quantitative Visual Acuity

SAE Serious Adverse Event/Serious Adverse Experience

SAP Statistical Analysis Plan SAS Statistical Analysis System

SD Standard Deviation

SOP Standard Operating Procedure

UADE Unanticipated Adverse Device Effect

USADE Unanticipated Serious Adverse Device Effect

VA Visual Acuity

#### 1. INTRODUCTION AND BACKGROUND

Cosmetic contact lenses can have patterns of varying size and opacities. When designing these cosmetic patterns, it is important to allow a sufficient clear area in the center of the lens optical zone so that the wearer's vision is not negatively impacted by the pattern.

In the current study, we will assess the objective visual performance of an investigation cosmetic soft contact lens compared to an approved cosmetic soft contact lens.

#### 1.1. Name and Descriptions of Investigational Products

This study will include two types of cosmetic contact lenses. The Control lens, 1-DAY ACUVUE® DEFINE® Radiant Sweet<sup>TM</sup> is an approved product, the Test, Etafilcon A Investigational Cosmetic Contact Lenses with PVP, is an investigational product. Further details about the test articles are found in Section 6 of this protocol.

#### 1.2. Intended Use of Investigational Products

The intended use of the investigational product is to correct vision. The investigational product contains a cosmetic pattern, so it also affects the visual appearance of the eye. During this non-dispensing study, each lens type will be worn for approximately 90 minutes.

#### 1.3. Summary of Findings from Nonclinical Studies

All previous pre-clinical findings were deemed satisfactory prior to proceeding with clinical trials on humans. For the most comprehensive nonclinical information regarding etafilcon A cosmetic contact lenses refer to the latest version of the Investigator's Brochure (Etafilcon A Investigational Limbal Ring Contact Lenses with polyvinylpyrrolidone [PVP]).

#### 1.4. Summary of Known Risks and Benefits to Human Subjects

The following risks/adverse events can be associated with wearing soft contact lenses in general:

- The eyes may burn, sting and/or itch.
- There may be a feeling of something in the eye (foreign body, scratched area).
- There may be the rare potential for some temporary impairment due to peripheral
  infiltrates, peripheral corneal ulcers and corneal erosion.
- There may be the rare potential for other physiological observations, such as local or generalized edema, corneal neovascularization, corneal staining, injection, tarsal abnormalities, iritis and conjunctivitis, some of which are clinically acceptable in low amounts.
- There may be excessive watering, unusual eye secretions, or redness of the eye.
- Poor visual acuity, blurred vision, rainbows or halos around objects, photo-phobia, or dry eyes may also occur if the lenses are worn continuously or for too long a time.
- Due to the reduction in light transmittance with cosmetically tinted lenses, some
  patients may experience visual symptoms while wearing the Study Contact
  Lenses. In addition, some patients may experience reduced peripheral awareness due
  to the opaque iris pattern.

There is no direct benefit to the subjects for participating in the study, although they will be able to try out marketed and investigational cosmetic contact lenses. The information from this study will aid if the further development and assessment of new potential cosmetic contact lenses.

For the most comprehensive clinical information regarding etafilcon A cosmetic contact lenses with PVP and the marketed contact lenses refer to the latest version of the Investigator's Brochure (Etafilcon A Investigational Limbal Ring Contact Lenses with PVP) and the package insert (APPENDIX C: PACKAGE INSERT (APPROVED PRODUCT).

# 1.5. Relevant Literature References and Prior Clinical Data Relevant to Proposed Clinical Study

There have been no serious or unanticipated adverse events and no loss of best correct VA reported in previous etafilcon A with PVP cosmetic contact lens clinical studies. There was one significant adverse event in \_\_\_\_\_\_, which was a small non-staining white corneal lesion. The site deemed this as not related to the study lenses as it was present prior to enrollment and stable at the final evaluation. See Clinical Study report for more information on this finding.

For the most comprehensive clinical information regarding etafilcon A cosmetic contact lenses with PVP and the marketed contact lenses refer to the latest version of the Investigator's Brochure (Etafilcon A Investigational Limbal Ring Contact Lenses with PVP) and the package insert (APPENDIX C: PACKAGE INSERT (APPROVED PRODUCT).

#### 2. STUDY OBJECTIVES, ENDPOINTS AND HYPOTHESES

#### 2.1. Objectives

Primary Objective

The primary objective of this study is to assess the objective vision of the study lenses at fitting.

**Exploratory Objective** 

Additional objectives include assessments of wavefront aberrometry, pupillometry, lens fit, subject reported ocular symptoms, and slit-lamp findings.

#### 2.2. Endpoints

Primary endpoints

Distance and Near Visual Acuity (logMAR)

LogMAR visual acuity will be assessed at distance (4 meters) and near (40 cm) using ETDRS Charts. This will be done using high and low contrast charts in bright illuminance conditions. Visual acuity will also be measured using high illumination and high contrast charts, while wearing neutral density goggles. See \_\_\_\_\_\_\_ for details regarding the collection of visual acuity (logMAR).

#### Quantitative Visual Acuity (qVA)

qVA will be measured under low room illumination (4 lux), low luminance, high contrast conditions with the M&S mesopic filter placed in front of the qVA monitor. Assessments will be made in OD and OU, seep Appendix E for additional details.

#### qCSF (CTP-2064)

Other Endpoints

#### Subjective Comfort and Vision

Comfort, vision and handling scores will be assessed using the Contact Lens User Experience (CLUE<sup>TM</sup>) questionnaire at lens fitting. CLUE is a validated patient-reported outcomes questionnaire to assess patient-experience attributes of soft, disposable contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Derived CLUE<sup>TM</sup> scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response with a range of 0-120. A 5-point increase in an average CLUE<sup>TM</sup> score translates into 10% shift in the distribution of scores for population of soft contact lens wearers<sup>5</sup>.

#### Wavefront aberrometry

Wavefront aberrometry will be assessed using a Visionix under dim lighting conditions (e.g. all lights off). Measurements will be taken as OS and OD, see Appendix F for additional details regarding the collection of wavefront aberrometry.

| Pupillometry | 7 |
|--------------|---|
|--------------|---|

#### Mechanical Lens fit

Lens fitting will be assessed in each eye using a slit-lamp post lens fitting; Lens fitting characteristics to be reported are:

- Lens Centration Grade
- Decentered Direction
- Limbal Exposure Grade
- Edge Lift (Present or Absent)
- Primary Gaze Movement Grade
- Upgaze Movement Grade
- Lens Tightness Grade (Push-up Test)
- Acceptable Fitting (yes/no)

#### Cosmetic Lens fit

Cosmetic lens fit assessment will be performed in each eye at post lens fitting by the investigator without the use of a slit-lamp at a distance of approximately 3 feet from the subject in:

- Primary Gaze
- Extreme Gaze (left and right)
- Extreme Up-gaze

#### Hula Hoop

If an investigator observes an unacceptable cosmetic lens fit in any gaze, a hula hoop assessment will be performed post lens fitting by the investigator without the use of a slit-lamp at a distance of approximately 3 feet from the subject in:

- Primary Gaze
- Extreme Gaze (left and right)
- Extreme Up-gaze

#### Ocular Physiology

Slit lamp findings will be assessed for each subject eye at baseline and the exit evaluation using the FDA Grading scale (Grade 0=None, Grade 1=Trace, Grade 2=Mild, Grade 3=Moderate, Grade 4=Severe). Slit lamp finding assessments include the following metrics:

- Corneal Infiltrates (Yes/No)
- Corneal Edema
- Corneal Neovascularization
- Corneal Neovascularization Location
- Corneal Staining
- Corneal Staining Location

- Conjunctival Injection
- Tarsal Abnormalities
- Other

See Appendices D and G for details about performing measurements of pupillometry, mechanical lens fit, cosmetic lens fit, hula hoop and ocular physiology.

#### 2.3. Hypotheses

Primary Hypotheses

Due to the exploratory nature of this study, there will be no planned hypotheses. Instead, descriptive summaries (i.e., tables and figures) of study endpoints will be provided for each lens type.

#### 3. TARGETED STUDY POPULATION

#### 3.1. General Characteristics

Subjects aged 18 to 39 years (inclusive) who are habitual soft contact lens wearers will be recruited for this clinical study. Subjects must meet all the inclusion and none of the exclusion criteria listed in Section 3.2. We will aim to enroll female subjects ages 18-29.

#### 3.2. Inclusion Criteria

Potential subjects must satisfy all of the following criteria to be enrolled in the study:

- The subject must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form
- 2. Appear able and willing to adhere to the instructions set forth in this clinical protocol
- 3. Subjects between 18 and 39 (inclusive) years of age at the time of screening
- 4. Be a current soft contact lens wearer in both eyes with a minimum of 6 hours/day and 5 days/week over the last month by self-report
- 5. The subject must be willing to be photographed and/or video-taped.

#### Eligibility after Baseline:

- 6. The subject's vertex corrected spherical equivalent distance refraction must be in the range of -1.00 D to -5.00 D (inclusive) in each eye
- 7. The subject's refractive cylinder must be less than or equal to 0.75 D (inclusive) in each eye
- 8. Have spherical best corrected visual acuity of 20/25 or better in each eye.

#### 3.3. Exclusion Criteria

Potential subjects who meet any of the following criteria will be excluded from participating in the study:

#### **Exclusion Criteria after Screening:**

- 1. Currently pregnant or lactating
- Any systemic disease (eg, Sjögren's Syndrome), allergies, infectious disease (eg, hepatitis, tuberculosis), contagious immunosuppressive diseases (eg, HIV), autoimmune disease (eg rheumatoid arthritis), or other diseases, by self-report, which are known to interfere with contact lens wear and/or participation in the study (at the investigators discretion)
- 3. Use of systemic medications (eg, chronic steroid use) that are known to interfere with contact lens wear (at the investigators discretion)
- Any previous, or planned (during the study) ocular surgery (eg, radial keratotomy, PRK, LASIK, etc.)
- Participation in any contact lens or lens care product clinical trial within seven (7) days prior to study enrollment
- Employee or family members of clinical site (eg, Investigator, Coordinator, Technician).

#### **Exclusion Criteria after Baseline**

- 7. Any ocular allergies, infections or other ocular abnormalities that are known to interfere with contact lens wear and/or participation in the study. This may include, but not be limited to entropion, ectropion, extrusions, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, aphakia, or corneal distortion (at the investigators discretion)
- Clinically significant (Grade 3 or 4 on FDA scale) tarsal abnormalities, bulbar injection, corneal edema, corneal vascularization, corneal staining, or any other abnormalities of the cornea which would contraindicate contact lens wear.

#### 3.4. Enrollment Strategy

Study subjects will be recruited from the Institution/clinical site's subject database and/or utilizing Independent Ethics Committee (IEC) or Institutional Review Board (IRB) approved materials by a market research company.

#### 4. STUDY DESIGN AND RATIONALE

#### 4.1. Description of Study Design

This is a single-site, single-visit, bilateral, randomized, controlled, 2 (lens)  $\times$  2 (period) crossover, non-dispensing study.

If a subject meets all eligibility criteria, they will be randomized to one of two lens wear sequences (Test/Control or Control/Test) is a bilateral fashion. Subjects will not be masked to the variant/pattern of the lenses due to visible differences; however, they will be masked to the lens brands. There will be a 5-minute washout period between study lenses.

#### 4.2. Study Design Rationale

Crossover designs are a well-established study design in which subjects are exposed to multiple treatments during different time periods. A 2X2 bilateral crossover design was considered to be the optimal design since the study period is relatively short the design can be cost effective and more efficient comparisons between treatments can be made than compared a parallel study since fewer subjects are required to achieve the same pre-specified statistical power. Each subject will act as their own control to reduce the influence of potential confounding factors such as age, gender and vision correction. Only a 5-minute washout between study lens wear will be implemented to help reduce any potential bias, since this is a non-dispensing study.

#### 4.3. Enrollment Target and Study Duration

Approximately 30 subjects ages 18 to 39 years (inclusive) who are habitual soft contact lens wearers will be enrolled in this single-visit clinical study with the goal of 25 subjects to complete. We will aim to enroll female subjects ages 18-29.

Enrollment is defined as execution of the informed consent form.

#### 5. TEST ARTICLE ALLOCATION AND MASKING

#### 5.1. Test Article Allocation

The study lenses will be worn in a bilateral and random fashion using a 2×2 crossover design. A computer-generated randomization scheme will be used to randomly assign subjects, in block of 2, to one of the two possible lens wear sequences: Test/Control or Control/Test. The random scheme will be generated using the PROC PLAN procedure from Statistical Analysis System (SAS) Software Version 9.4 or higher (SAS Institute, Cary, NC).

The study site must follow the randomization scheme provided and complete enrollment per the randomization list and not pre-select or assign subjects. The randomized assignment of subjects will be performed at the first visit prior to the first fitting. The following must have occurred prior to randomization:

- Informed consent has been obtained
- Subject meets all the inclusion / exclusion criteria
- Subject history and baseline information has been collected.

#### 5.2. Masking

Due to visible print differences, subjects and investigators will be aware of the different patterns/variants of the investigational product. However, subjects will be masked to the lens brand to prevent bias during the lens discussions.

Under normal circumstances, the mask should not be broken until all subjects have completed the study and the database is finalized. Otherwise, the mask should be broken only if specific emergency treatment/course of action would be dictated by knowing the treatment status of the subject. In such cases, the Investigator may, in an emergency, contact the medical monitor. In the event the mask is broken the Sponsor must be informed as soon as possible. The date, time, and reason for the unmasking must be documented in the subject record. The Investigator is also advised not to reveal the study treatment assignment to the clinical site or Sponsor personnel.

Subjects who have had their treatment assignment unmasked are expected to return for all remaining scheduled evaluations. Subjects who are discontinued may be replaced.

#### 5.3. Procedures for Maintaining and Breaking the Masking

The Clinical Supply Unit will generate a unique code for all study lenses. Marketed products and investigational lenses will have nearly identical labels, differing only in the product specifications and lens code, to maintain masking. Subjects will be dispensed lenses by the lens code in accordance with the randomization scheme provided by the study statistician.

The test articles mask shall not be broken unless information concerning the lens type is necessary for the urgent medical treatment of a subject. The Sponsor must be notified before the mask is broken.

When dispensing test articles, the following steps should be followed to maintain randomization codes:

- Investigator or designee (documented on the Delegation Log) will consult the lens fitting schedule/randomization scheme to obtain the test article assignment for that subject prior to dispensing.
- Investigator or designee will record the subject's number on the appropriate line of the randomization scheme.
- 3. Investigator or designee will pull the appropriate test articles from the study supply. All test articles that are opened, whether dispensed (placed/fit on eye or dispensed outside the clinical site) or not, must be recorded on the Test Article Accountability Log in the "Dispensed" section.

#### 6. STUDY INTERVENTION

#### 6.1. Identity of Test Articles

The following contact lenses will be used in this study:

Table 1: Test Articles

| | Control | Test |
|---|---|---|
| Name | 1-DAY ACUVUE <sup>®</sup> DEFINE <sup>®</sup><br>Radiant Sweet™ | Etafilcon A with PVP with cosmetic pattern Green |
| Manufacturer | Johnson & Johnson | Johnson & Johnson |
| Lens Material | Etafilcon A | Etafilcon A |
| Nominal Base Curve @ 22°C | 8.5 mm | 8.5 mm |
| Nominal Diameter @ 22°C | 14.2 mm | 14.2 mm |
| Nominal Distance<br>Powers (D) | -1.00 to -5.00 D | -1.00 to -5.00 D |
| Modality in Current<br>Study | Daily | Daily |
| Replacement<br>Frequency | Daily | Daily |
| Packaging Form (vial, blister, etc.) | Blister | Blister |

Each subject will wear approximately 2 of each lens type.

#### 6.2. Ancillary Supplies/Products

The following solutions will be used in this study:

Sensitive Eyes Plus (Bausch & Lomb) or country-specific alternative approved by the sponsor, FluStrips (Contacare) or country-specific alternative approved by the sponsor, and Tears Naturale Free (Alcon) or country-specific alternative approved by the sponsor.

Table 2: Ancillary Supplies

| | | Solution | |
|---|---|---|---|
| Solution Name/Description | Sensitive Eyes<br>plus Saline (or<br>other sponsor-<br>approved<br>product) | Tears Naturale<br>Free (or other<br>sponsor-<br>approved<br>product) | FluStrips Fluorescein (or other sponsor- approved product) |
| Manufacturer | Bausch & Lomb | Alcon | Contacare<br>Ophthalmics<br>Diagnostics<br>(EOU) |
| Preservative | None | None | None |
| Other distinguishing items (dye, packaging, approval status, etc. | NA | NA | D&C Yellow No.<br>8, 0.6 mg |

#### 6.3. Administration of Test Articles

Test articles will be dispensed to subjects meeting all eligibility requirements, including any dispensing requirements set forth in this clinical protocol. Subjects will be dispensed an adequate supply of test articles to complete the study. Lost or damaged test articles may be replaced at the discretion of the Investigator and/or the Sponsor.

#### 6.4. Packaging and Labeling

The test articles will be over-labeled to mask the subject/Investigators to the identity of the lens. The labels will meet the country-specific labeling guidelines for clinical studies involving investigational contact lenses. The test articles will be in plastic bags as the secondary packaging form.

The sample study label is shown below:

CPL-Label- A

#### 6.5. Storage Conditions

Test articles will be maintained at ambient temperatures at the clinical site. Test articles must be kept under secure conditions.

#### 6.6. Collection and Storage of Samples

No samples will be collected as part of the study procedures.

When possible, any lens or test article associated with an Adverse Events and/or a Product Quality Complaint must be retained and stored in a glass vial with moderate solution pending directions from the sponsor for potential return back to JJVC.

#### 6.7. Accountability of Test Articles

JJVC will provide the Investigator with sufficient quantities of study articles and supplies to complete the investigation. The Investigator is asked to retain all lens shipment documentation for the test article accountability records.

Test articles must be kept in a locked storage cabinet, accessible only to those assigned by the Investigator for dispensing. The Investigator may delegate this activity to authorized study site personnel listed on the Site Delegation Log. All test articles must be accounted. This includes:

- 1. What was dispensed for the subject for trial fitting, to wear out of the office, or issued for the subject to replace appropriately between visits.
- 2. What was returned to the Investigator unused, including expired or malfunctioning product.
- 3. The number and reason for unplanned replacements.

The Investigator will collect all unused test articles from the subjects at the end of the subject's participation. Subject returned unused test articles must be separated from the clinical study inventory of un-dispensed test articles and must be labeled with the subject number and date of return. Following final reconciliation of test articles by the monitor, the Investigator or monitor will return all unused test articles to JJVC.

| Î | Site | Instructions | for | Test | Article | Receipt | and | Test | Article |
|---|---|---|---|---|---|---|---|---|---|

#### 7. STUDY EVALUATIONS

#### 7.1. Time and Event Schedule

Table 3: Time and Events

| Event | Visit 1:<br>Screening<br>Baseline | Visit 1:<br>Treatment 1 | Visit 1:<br>Treatment 2 |
|---|---|---|---|
| Time point | | Day 0 | |
| Visit Duration | | 4.5 hours | |
| Statement of Informed Consent | X | | |
| Demographics | X | | |
| Inclusion/Exclusion Criteria | X | | |
| Medical History | X | | |
| Concomitant Medication | X | | |
| Habitual Lens Information | X | | 3 |
| Subject Reported Ocular Symptoms | | X | X |
| Entrance Visual Acuity | X | | |
| Subjective Sphero-Cylindrical Refraction | X | | |
| Subjective Best Sphere Refraction | X | | |
| Pupillometry | | X | |
| Entrance Slit Lamp Exam | X | | |
| Lens Assignment | | X | X |
| Lens Insertion | | X | X |

| Event | Visit 1:<br>Screening | Visit 1:<br>Treatment 1 | Visit 1:<br>Treatment 2 |
|---|---|---|---|
| | Baseline | | |
| Time point | | Day 0 | |
| Visit Duration | | 4.5 hours | |
| Lens Settling | | X | X |
| Over Refraction | | X | X |
| Visual experience | | X | X |
| PRO Post Fit Questionnaire | | X | X |
| logMAR Visual performance (distance and near) | | X | X |
| qCSF | 2 | X | X |
| qVA | | X | X |
| Wavefront aberrometry | X | X | X |
| Cosmetic Lens Fit (without slit-lamp) | | X | X |
| Hula Hoop Evaluation (without slit-lamp) | | X | X |
| Mechanical Lens Fit Assessment | 4 | X | X |
| Exit Slit Lamp Exam | | | X |
| Exit Snellen Distance VA | 2 | | X |
| Study Completion/ Adverse Event Review | | | X |
| Final Exam Form and Investigator Signature | | | X |

### 7.2. Detailed Study Procedures

#### VISIT 1

The subject must attend the visit wearing their habitual spectacles (where applicable).

| | | Visit 1: Screening | 141 |
|---|---|---|---|
| Step | Procedure | Details | |
| 1.1 | Statement of<br>Informed Consent | Each subject must read, understand, and sign the Statement of Informed Consent before being enrolled into the study. The Principal Investigator or his/her designee conducting the informed consent discussion must also sign the consent form. Note: The subject must be provided a signed copy of this document. | |
| 1.2 | Demographics | Record the subject's year of birth, gender, race and ethnicity. | |
| 1.3 | Medical History and<br>Concomitant<br>Medications | Questions regarding the subjects' medical history and concomitant medications. | |
| 1.4 | Habitual Lenses | Questions regarding the subject's habitual lens type, parameters, wear schedule and duration. | |

| 1.5 | Eligibility after<br>Screening | All responses to Screening Inclusion Criteria questions must be answered "yes" and all responses to Exclusion Criteria must be answered "no" for the subject to be considered eligible. |
|---|---|---|
| | | If subject is deemed to be ineligible after screening, proceed to Final Evaluation and complete Subject Disposition. Visual Acuity, Refraction and Biomicroscopy forms are not required. |

| | | Visit 1: Baseline |
|---|---|---|
| Step | Procedure | Details |
| 1.6 | Entrance Visual<br>Acuity | Record the distance Snellen visual acuity (OD, OS, and OU) to the nearest letter with their habitual spectacles (where applicable). Subjects must read the smallest line until at least 50% of the letters are read incorrectly. |
| 1.7 | Subjective Sphero-<br>cylindrical<br>Refraction | Complete subjective spherocylindrical refraction and record the resultant distance visual acuity (OD, OS and OU) to the nearest letter. |
| 1.8 | Subjective Best<br>Sphere Refraction | Perform subjective best sphere refraction with a phoropter (adopt the maximum plus to maximum visual acuity (MPMVA) approach and use the duo-chrome test for binocular balancing) and record the best corrected distance visual acuity (OD, OS, OU) to the nearest letter. Note: The endpoint criterion for the duo-chrome test is the lens power at which the red and green sides of the chart appear to be equally distinct. However, if the subject's response changes from "red" to "green" with only a 0.25D change in power and no report that the two sides appear to be equally sharp, the refraction endpoint should be the lens power that leave the red chart sharper. Note 2: The subject's optimal vertexed spherical equivalent distance correction must be between -1.00D and -5.00D. |

| 1.9 | Visionix VX118 | Measure the wavefront for each eye with the | |
|---|---|---|---|
| | Wavefront (if | Visionix VX118 instrument (using WF | |
| | available) | mode) in dim room illumination. | |
| | | On the Coeff. Aberr. tab, select RL display | |
| | | and Night mode, then record the pupil size (in | |
| | | mm), HOA (in microns) and the Sph. Aberr. | |
| | | (in microns) for each eye. | |
| 1.10 | Slit Lamp Findings | FDA Slit Lamp Classification Scale will be | |
| | | used to grade the findings and determine | - Table |
| | | eligibility. | |
| | | If any of these slit lamp findings are Grade 3 | |
| | | or higher, the subject may not continue at this | |
| | | time, but may return up to one additional time<br>to determine eligibility. If discontinued a | |
| | | final examination must be completed. | |
| | | imar examination must be completed. | |
| | | If the clearance of the fluorescein needs to be | |
| | | expedited, preservative-free rewetting drops | |
| | | or saline may be instilled. | |
| 1.11 | Eligibility after | All responses to Inclusion Criteria questions | |
| 120000000000000000000000000000000000000 | Baseline | must be answered "yes" and all responses to | |
| | | Exclusion Criteria questions must be | |
| | | answered "no" for the subject to be | |
| | | considered eligible. | |

| | | Visit 1: Treatment 1 Lens Fitting |
|---|---|---|
| Step | Procedure | Details |
| 1.12 | Lens Selection | Assign the study lens based on the randomization scheme. Select the contact lens power based on subjective best sphere refraction. |
| 1.13 | Lens Insertion | The Investigator or the subject inserts the study lenses. Record the time of lens insertion. Check for lens damage under the slit lamp before proceeding with lens settling. Replace damaged lenses if applicable. Note: Designated site staff should observe the insertion process. If it appears that the subject attempts to insert a lens that is "inside-out", they should interfere to avoid incorrect insertion. Note 2: If the lens moves excessively on the eye after insertion, ask the subject to remove |

| | | the lens, confirm lens is not inverted (correct | |
|---|---|---|---|
| | · ~ | if it is is) and reinsert. | |
| 1.14 | Lens Settling | Allow the study lenses to settle for a | |
| 1.15 | C 1: · | minimum of 5 minutes. | |
| 1.15 | Subjective Best | Perform subjective best sphere refraction over | |
| | Sphere Over<br>Refraction | the study lenses with a phoropter (adopt the | |
| | Refraction | maximum plus to maximum visual acuity | |
| | | (MPMVA) approach and use the duo-chrome test for binocular balancing) and record the | |
| | | best corrected distance visual acuity to the | |
| | | nearest letter (OD, OS, OU). | |
| 1.16 | Lens Power | Adjust the lens power if the subject's best | |
| | Modification (if | sphere over-refraction is not plano. | |
| | applicable) | For each power modification, repeat steps | |
| | | (1.13 to 1.16). | |
| | | Only two power modifications per eye are | |
| 1.17 | G 1: + D + 1 | allowed. | |
| 1.17 | Subject Reported | Subjects will respond to a verbal open-ended | |
| 1.18 | Ocular Symptoms Visual Experience | symptoms questionnaire. Subject will spend approximately 20 minutes | |
| 1.18 | visual Experience | experiencing vision. During this time please | |
| | | instruct subject to look outside (windows or | - |
| | | physically walk outside), use electronic | |
| | | device (phone, computer), read magazine | |
| | | print, and experience dim room illumination | |
| | | for tasks. A member of the clinical site must | |
| | | accompany the subject at all times if outside | |
| | | the clinic area. | |
| 1.19 | Post-Fit | The subject will respond to the CLUE/PRO | |
| | Questionnaire | Post-Fit Questionnaire. | |
| 1.20 | Distance ETDDC | Don | |
| 1.20 | Distance ETDRS LogMAR Visual | Per please confirm room illuminance and chart luminance | |
| | Acuity- High | acceptable ranges for both high/low contrast | |
| | illumination | visual acuity testing. | |
| | III WIII III WIII VII | ribual acuity testing. | |
| | | 1. Under high illumination and high chart | |
| | | luminance, record the distance (4 meter) | |
| | | ETDRS high contrast visual acuity OD | |
| | | (HC1) and OU (HC2). | |
| | | 2. Under high illumination and high chart | |
| | | luminance, record the distance (4 meter) | |
| | | ETDRS low contrast visual acuity OD | |
| | | (LC1) and OU (LC2). | |
| L | l . | l | |

| | | Letter-by-letter results will be recorded into<br>the electronic data capture form, which will<br>calculate the visual performance score for each<br>chart read. |
|---|---|---|
| 1.21 | Near logMAR<br>Visual Acuity- High<br>illumination | Per please confirm room illuminance and chart luminance acceptable ranges for both high/low contrast visual acuity testing. |
| | | 1. Under high illumination and high chart luminance, record the near (40 cm) low contrast visual acuity OD and OU (once each). |
| | | Letter-by-letter results will be recorded into<br>the electronic data capture form, which will<br>calculate the visual performance score for each<br>chart read. |
| | | Regarding Near logMAR VA: the room illumination will be >400 lux for all testing Regarding the Near logMAR VA |
| | | Reference to verification chart and room illuminance is not applicable |
| 1.22 | Distance ETDRS LogMAR Visual Acuity- with googles | Per please confirm room illuminance and chart luminance acceptable ranges for both high/low contrast visual acuity testing. |
| | | 1. With the goggles on, under high illumination and chart luminance, record the distance (4 meter) ETDRS high contrast visual acuity OD (HC3) and OU (HC4). Allow subject to adjust to dim condition for 3 minutes. |
| | | Letter-by-letter results will be recorded into<br>the electronic data capture form, which will<br>calculate the visual performance score for<br>each chart read. |
| 1.23 | Near logMAR<br>Visual Acuity- with<br>goggles | Per please confirm room illuminance and chart luminance acceptable ranges for both high/low contrast visual acuity testing. |

| | | 1. With the goggles on, under high illumination and chart luminance, record the near (40 cm) high contrast visual acuity OD and OU (once each). Allow subject to adjust to dim condition for 3 minutes (if not already adjusted) |
|---|---|---|
| | | Letter-by-letter results will be recorded into the electronic data capture form, which will calculate the visual performance score for each chart read. Regarding Near logMAR VA: the room illumination will be >400 lux for all testing Regarding the Near logMAR VA |
| | | Reference to verification chart and room |
| 1.24 | Quick Contrast | illuminance is not applicable Conduct OD and OU with 25 trials. |
| 1.27 | Sensitivity Function (qCSF) | Conduct OD and OO with 23 trials. |
| 1.25 | Pupillometry | With the subject facing the qCSF monitor and under the same dim light conditions that qCSF was measured, take 3 measurements of the pupil size of the subjects OD and OS with the pupillometer. |
| 1.26 | Quantitative Visual<br>Acuity (qVA) | A demonstration trial must be performed prior to any data collection |
| | | Complete the qVA measurement of the OD and OU utilizing the following qVA configurations: • Number of rows: 15 • Stimulus duration: 3 seconds • Test Distance: 4 meters • Under low room illumination (4 lux), low luminance, high contrast conditions (with the M&S mesopic filter placed in front of the qVA monitor) |
| | | Allow subject to adjust to dim condition for 3 minutes (if not already adjusted) |
| | | EDC to record qVAt (threshold) in logMAR and qVAr (range) in lines |

| 1.27 | Visionix VX118 Wavefront (if available) Cosmetic Lens Fit Assessment (without slit-lamp) | Measure the wavefront for each eye with the Visionix VX118 instrument (using WF mode) in dim room illumination. On the Coeff. Aberr. tab, select RL display and Night mode, then record the pupil size (in mm), HOA (in microns) and the Sph. Aberr. (in microns) for each eye. The Cosmetic Lens Assessment will be assessed by the investigator (without slitlamp) in primary gaze and extreme gaze (right, left, and upgaze) at a normal conversation distance (approximately three |
|---|---|---|
| 1.29 | Hula Hoop Assessment (without slit-lamp) *if unacceptable cosmetic lens fit in any gaze* | (3) feet away from the subject). If there is an unacceptable cosmetic fit in any gaze, the Hula Hoop Assessment will be assessed by the investigator (without slitlamp) in primary gaze and extreme gaze (right, left, and upgaze) at a normal conversation distance (approximately three (3) feet away from the subject). |
| 1.30 | Subjective Lens Fit<br>Assessment | Evaluate overall lens fit acceptance (acceptable or unacceptable) based on centration, movement and other fitting characteristics. An unacceptable fit is deemed by one of the following criteria: Iimbal exposure at primary gaze or with extreme eye movement; edge lift; excessive movement in primary and up gaze; or insufficient movement in all three of the following conditions: primary gaze, up gaze, and Josephson push up. If the fit is unacceptable, the subject can continue with the study. |
| 1.31 | Photographs/Videos | Photographs/Videos of the lenses on eye may be taken if there is an unacceptable cosmetic or mechanic lens fit. |
| 1.32 | Remove lenses | Have subject remove lenses. Worn lenses can be discarded. |
| 1.33 | Washout | There will be a 5-minute washout between lenses |

| | Visit 1: Treatment 2 Lens Fitting | |
|---|---|---|
| Step | Procedure | Details |
| 1.34 | Lens Selection | Assign the study lens based on the randomization scheme. Select the contact lens power based on subjective best sphere refraction. |
| 1.35 | Lens Insertion | The Investigator or the subject inserts the study lenses. Record the time of lens insertion. Check for lens damage under the slit lamp before proceeding with lens settling. Replace damaged lenses if applicable. Note: Designated site staff should observe the insertion process. If it appears that the subject attempts to insert a lens that is "inside-out", they should interfere to avoid incorrect insertion. |
| | | Note 2: If the lens moves excessively on the eye after insertion, ask the subject to remove the lens, confirm lens is not inverted (correct if it is is) and reinsert. |
| 1.36 | Lens Settling | Allow the study lenses to settle for a minimum of 5 minutes. |
| 1.37 | Subjective Best<br>Sphere Over<br>Refraction | Perform subjective best sphere refraction over<br>the study lenses with a phoropter (adopt the<br>maximum plus to maximum visual acuity<br>(MPMVA) approach and use the duo-chrome<br>test for binocular balancing) and record the<br>best corrected distance visual acuity to the<br>nearest letter (OD, OS, OU). |
| 1.38 | Lens Power<br>Modification (if<br>applicable) | Adjust the lens power if the subject's best sphere over-refraction is not plano. For each power modification, repeat steps (1.35 to 1.38). Only two power modifications per eye are allowed. |
| 1.39 | Subject Reported<br>Ocular Symptoms | Subjects will respond to a verbal open-ended symptoms questionnaire. |

| 1.40 | Visual Experience | Subject will spend approximately 20 minutes experiencing vision. During this time please instruct subject to look outside (windows or physically walk outside), use electronic device (phone, computer), read magazine print, and experience dim room illumination for tasks. A member of the clinical site must accompany the subject at all times if outside the clinic area. |
|---|---|---|
| 1.41 | Post-Fit<br>Questionnaire | The subject will respond to the CLUE/PRO Post-Fit Questionnaire. |
| 1.42 | Distance ETDRS logMAR Visual Acuity- High illumination | Per please confirm room illuminance and chart luminance acceptable ranges for both high/low contrast visual acuity testing. |
| | | 3. Under high illumination and high chart luminance, record the distance (4 meter) ETDRS high contrast visual acuity OD (HC1) and OU (HC2). |
| | | 4. Under high illumination and high chart luminance, record the distance (4 meter) ETDRS low contrast visual acuity OD (LC1) and OU (LC2). |
| | | Letter-by-letter results will be recorded into<br>the electronic data capture form, which will<br>calculate the visual performance score for each<br>chart read. |
| 1.43 | Near logMAR Visual Acuity- High illumination | Per please confirm room illuminance and chart luminance acceptable ranges for both high/low contrast visual acuity testing. |
| | | 2. Under high illumination and high chart luminance, record the near (40 cm) low contrast visual acuity OD and OU (once each). |
| | | Letter-by-letter results will be recorded into<br>the electronic data capture form, which will<br>calculate the visual performance score for each<br>chart read. |

| | | Dogarding Near logMAD VA. |
|---|---|---|
| | | Regarding Near logMAR VA:<br>the room illumination will be >400 lux for all |
| | | testing |
| | | Regarding the Near logMAR VA |
| | | Reference to verification chart and room |
| | | illuminance is not applicable |
| 1.44 | Distance ETDRS | Per , please confirm |
| | LogMAR Visual | room illuminance and chart luminance |
| | Acuity- with googles | acceptable ranges for both high/low contrast |
| | | visual acuity testing. |
| | | 2. With the goggles on, under high |
| | | illumination and chart luminance, |
| | | record the distance (4 meter) ETDRS |
| | | high contrast visual acuity OD (HC3) |
| | | and OU (HC4). Allow subject to adjust |
| | | to dim condition for 3 minutes. |
| | | Letter-by-letter results will be recorded into |
| | | the electronic data capture form, which will |
| | | calculate the visual performance score for |
| | | each chart read. |
| 1.45 | Near logMAR | Per please confirm room |
| | Visual Acuity- with | illuminance and chart luminance acceptable |
| | goggles | ranges for both high/low contrast visual acuity |
| | 8 88 | testing. |
| | | 5 |
| | | 2. With the goggles on, under high |
| | | illumination and chart luminance, |
| | | record the near (40 cm) high contrast |
| | | visual acuity OD and OU (once each). |
| | | • |
| | | Allow subject to adjust to dim condition |
| | | for 3 minutes (if not already adjusted) |
| | | Letter-by-letter results will be recorded into |
| | | the electronic data capture form, which will |
| | | calculate the visual performance score for each |
| | | chart read. |
| | | Regarding Near logMAR VA: |
| | | the room illumination will be >400 lux for all |
| | | testing |
| | | Regarding the Near logMAR VA |
| | | regarding the rear logivitals via |
| | | Reference to verification chart and room |
| 1 | | illuminance is not applicable |

| 1.46 | Quick Contrast Sensitivity Function (qCSF) | Conduct OD and OU with 25 trials. |
|---|---|---|
| 1.47 | Quantitative Visual<br>Acuity (qVA) | A demonstration trial must be performed prior to any data collection Complete the qVA measurement of the OD and OU utilizing the following qVA configurations: Number of rows: 15 Stimulus duration: 3 seconds Test Distance: 4 meters Under low room illumination (4 lux), low luminance, high contrast conditions (with the M&S mesopic filter placed in front of the qVA monitor) Allow subject to adjust to dim condition for 3 minutes (if not already adjusted). EDC to record qVAt (threshold) in logMAR and qVAr (range) in lines |
| 1.48 | Visionix VX118<br>Wavefront (if<br>available) | Measure the wavefront for each eye with the Visionix VX118 instrument (using WF mode) in dim room illumination. On the Coeff. Aberr. tab, select RL display and Night mode, then record the pupil size (in mm), HOA (in microns) and the Sph. Aberr. (in microns) for each eye. |
| 1.49 | Cosmetic Lens Fit<br>Assessment (without<br>slit-lamp) | The Cosmetic Lens Assessment will be assessed by the investigator (without slit-lamp) in primary gaze and extreme gaze (right, left, and upgaze) at a normal conversation distance (approximately three (3) feet away from the subject). |
| 1.50 | Hula Hoop Assessment (without slit-lamp) *if unacceptable cosmetic lens fit in any gaze* | If there is an unacceptable cosmetic fit in any gaze, the Hula Hoop Assessment will be assessed by the investigator (without slit-lamp) in primary gaze and extreme gaze (right, left, and upgaze) at a normal conversation distance (approximately three (3) feet away from the subject). |
| 1.51 | Subjective Lens Fit<br>Assessment | Evaluate overall lens fit acceptance (acceptable or unacceptable) based on centration, movement and other fitting characteristics. An unacceptable fit is deemed by one of the following criteria: Imbal exposure at primary gaze or with extreme eye movement; edge lift; excessive movement in primary and up gaze; or insufficient movement in all three of the following conditions: primary gaze, up gaze, and Josephson push up. If the fit is unacceptable, the subject can continue with the study. |
|---|---|---|
| 1.52 | Photographs/Videos | Photographs/Videos of the lenses on eye may be taken if there is an unacceptable cosmetic or mechanic lens fit. |
| 1.53 | Remove lenses | Have subject remove lenses. Worn lenses can be discarded. |

## FINAL EVALUATION

The final evaluation will ordinarily take place immediately following the last scheduled follow-up visit per the study protocol. It may also take place at any point the subject discontinues the study or is terminated from the study.

| Final Evaluation | | |
|---|---|---|
| Step | Procedure | Details |
| F.1 | Final Exam Form | Indicate if the subject completed the study successfully. If subject discontinued from the study, indicate the reason. |
| F.2 | Exit Slit Lamp<br>Biomicroscopy | FDA Slit Lamp Classification Scale will be used to grade the findings. If no slit lamp finding is noted on the EDC form it is considered as a zero "0" Grade for all observations listed. After the slit lamp examination, at the discretion of the Investigator, rinse the subject's eyes thoroughly with preservative-free saline. |

| Final Evaluation | | |
|---|---|---|
| Step | Procedure | Details |
| F.3 | Exit Visual Acuity | Record the distance Snellen visual acuity (OD, OS, and OU) to the nearest letter with their habitual spectacles (where applicable). Subjects must read the smallest line until at least 50% of the letters are read incorrectly. |

#### 7.3. Unscheduled Visits

If, during the investigation, a subject requires an unscheduled visit to the clinical site, the following information will be collected as appropriate:

- Chief complaint prompting the visit. If the reason is an adverse event, the applicable eCRF for the adverse event must be completed and subject record completed as appropriate.
- Date and time of the visit and all procedures completed at the unscheduled visit.
- Review of adverse event and concomitant medications.
- Slit lamp findings (using the Slit Lamp Classification Scale).

If the Investigator withdraws a subject from the study, the final study visit case report forms must be completed indicating the reason(s) why the subject was withdrawn. The subject record must be completed documenting the date and primary reason for withdrawal and the study CRA notified.

Any ocular and non-ocular Adverse Events that are ongoing at the time of the study visit will be followed by the Investigator, within licensure, until they have resolved, returned to pretreatment status, stabilized, or been satisfactorily explained. If further treatment i.e., beyond licensure is required, the subject will be referred to the appropriate health care provider.

The following information will be collected during an unscheduled visit as appropriate.

| Unscheduled Visit | | |
|---|---|---|
| Step | Procedure | Details |
| U.1 | Chief Complaints | Record the subject's chief complaints for reasons for the unscheduled visit. |
| U.2 | Adverse Events and<br>Concomitant<br>Medications Review | Review any changes to the subject's medical history or concomitant medications from the previous study visit. Record any changes, and any adverse events. |
| U.3 | Entrance VA | Record the entrance distance visual acuity (OD, OS and OU) to the nearest letter. |

| | Unscheduled Visit | |
|---|---|---|
| Step | Procedure | Details |
| U.4 | Subjective Sphero-<br>cylindrical<br>Refraction | Perform bare-eye subjective spherocylindrical refraction with a phoropter (adopt the maximum plus to maximum visual acuity (MPMVA) approach and use the duo-chrome test for binocular balancing) and record the best corrected distance visual acuity to the nearest letter (OD, OS, and OU). |
| U.5 | Slit Lamp<br>Biomicroscopy | FDA Slit Lamp Classification Scale will be used to grade the findings. If the clearance of the fluorescein needs to be expedited, preservative-free rewetting drops may be instilled. |
| U.6 | Exit Visual Acuity | Record the subject's exit distance visual acuity (OD, OS, and OU) to the nearest letter. |

## 7.4. Laboratory Procedures

Not Applicable

#### 8. SUBJECTS COMPLETION/WITHDRAWAL

## 8.1. Completion Criteria

Subjects are considered to have completed the study if they:

- provided informed consent and/or assent;
- they are eligible;
- Completed all study visits;
  - Have not withdrawn/discontinued from the study for any reason described in Section 8.2

#### 8.2. Withdrawal/Discontinuation from the Study

A subject will be withdrawn from the study for any of the following reasons:

- Subject death during the study period
- Subject withdrawal of consent and/or assent
- Subject not compliant to protocol
- Subject lost to follow-up
- Subject no longer meets eligibility criteria (eg the subject becomes pregnant)
- Subject develops significant or serious adverse events causing discontinuation of study lens wear
- Subjects who have experienced a Corneal Infiltrative Event (CIE)
- Investigator's clinical judgment regarding the subject safety reasons (that it is in the best interest of the subject to stop treatment)

For discontinued subjects, the Investigator will:

- Complete the current visit (scheduled or unscheduled)
- Complete the Final Evaluation, indicating the reason that the subject was discontinued from the study
- Record the spherocylindrical refraction with best corrected distance visual acuity, as appropriate
- Collect used test article(s) (worn or brought to the visit) from the subject and discard them, unless otherwise stated in Section 7.2
- Collect all unused test article(s) from the subject

An additional subject may be enrolled if a subject discontinues from the study prematurely.

In cases where a subject is lost to follow-up, every possible effort must be made to contact the subject and determine the reason for discontinuation/withdrawal. The measures taken to follow up must be documented including two written attempts and a certified letter (or equivalent) as the final attempt.

#### 9. PRE-STUDY AND CONCOMITANT INTERVENTION/MEDICATION

Concomitant medications will be documented during screening and updated during the study. Disallowed medications for this study include: None Concomitant therapies that are disallowed include: None

## 9.1. Systemic Medications

Due to the non-dispensing, single visit nature of the study and endpoints being assessed, systemic medications will be allowed provided they did not interfere with contact lens wear, which will be at the discretion of the investigator.

Disallowed systemic medications - Not applicable

#### 10. DEVIATIONS FROM THE PROTOCOL

Investigator will notify study sponsor upon identification of a protocol deviation. Protocol deviations must be reported to the sponsor within 24 hours after discovery of the protocol deviation. The Investigator will report deviations per IRB/IEC requirements. All deviations will be tracked and corrective actions implemented as appropriate.

If it becomes necessary for the Investigator to implement a deviation in order to eliminate an immediate hazard to the trial subject, the Investigator may implement the deviation immediately without notification to the sponsor. Within 24 hours after the implemented deviation, the Investigator must notify and provide the rationale to the Sponsor and, as required, the IEC/IRB.

If the deviation potentially impacts the safety of patient or changes the technical integrity of the study then it must be reported to IEC/IRB. This is a "Major Deviation".

Minor deviations have no substantive effect on patient safety or technical integrity of the study. They are often logistical in nature. The informed consent must also not be contradicted by the deviation.

Protocol waivers are prohibited

#### 11. STUDY TERMINATION

The occurrence of one or more Unanticipated Serious Adverse Device Effect (USADE), or any SAE where the relationship to study agent cannot be ruled out, may result in stopping further dispensing of test article. In the event of a USADE or SAE, the Sponsor may unmask the treatment regimen for the subject(s) and will discuss this with the Investigator before any further subjects are enrolled.

The Sponsor will determine when a study will be stopped. The Principal Investigator always has the discretion to initiate stopping the study based on patient safety or if information indicates the study's results are compromised.

JJVC reserves the right to terminate the study at any time for any reason. Additionally, the IEC/IRB reserves the right to terminate the study if an unreasonable risk is determined. The study can be terminated by the Principal Investigator at the individual clinical site due to specific clinical observations, if in their opinion, after a discussion with JJVC, it is determined that it would be unwise to continue at the clinical site.

JJVC (and the IEC/IRB and DMC, if applicable) will evaluate all adverse events. If it is determined that an adverse event presents an unreasonable risk, the investigation, or that part of the investigation presenting the risk, will be terminated as soon as possible.

Should the study be terminated (either prematurely or as scheduled), the Investigator will notify the IEC/IRB and Regulatory Authority as required by local regulatory requirements.

## 12. PROCEDURE FOR HANDLING PRODUCT QUALITY COMPLAINTS

A Product Quality Complaint (PQC) refers to any written, electronic, or oral communication that alleges deficiencies related to the identity, quality, durability, reliability, safety, effectiveness or performance of test articles after they have been released for clinical trial use.

Potential complaints may come from a variety of sources including but not limited to subjects, clinical research associates (CRA), clinical operations managers (COM), medical monitors, and site personnel, etc. The following are not considered product quality complaints:

• Subject satisfaction inquiries reported via "Subjective Questionnaires" and "Patient Reported Outcomes (PRO)."

- Clinical test articles that are stored improperly or damaged after receipt at the investigational site.
- Lens replacements that occur due to drops/fall-outs.
- Damage deemed by clinicians or clinical staff to be caused by handling by the user, and not indicative of a quality deficiency (i.e. tears, rips, etc.), only in situations where there is no deficiency alleged by the subject.

Within 24 hours of site personnel becoming aware that a PQC has occurred, the PQC must be recorded in the EDC system, which will trigger an automatic email notification to the appropriate COM/CRA and Clinical QA representative. In cases where the EDC system in use is not configured to send automatic notifications or when an EDC system is not used, the COM/CRA is responsible for notifying Clinical QA upon discovery that a PQC has occurred.

Upon receipt of the EDC notification, the COM/CRA will contact the study site to collect additional information which will include:

- Date the complaint was received/recorded in the EDC System (Date of Sponsor Awareness).
- Who received the complaint.
- Study number.
- Clinical site information (contact name, site ID, telephone number).
- Lot number(s).
- Unique Subject Identifier(s).
- Indication of who first observed complaint (site personnel or subject).
- OD/OS indication, along with whether the lens was inserted.
- Any related AE number if applicable.
- Detailed complaint description (scheduled/unscheduled visit, wear time, symptoms, resolution of symptoms, etc.).
- Eye Care Provider objective (slit lamp) findings if applicable.
- Confirmation of product availability for return (and tracking information, if available), or rationale if product is not available for return (for test article return instructions).

Once a complaint is received, it will be assessed by the COM, CRA, or trained site personnel to determine if it is an Adverse Event/Serious Adverse Event (AE/SAE). If the complaint results in an AE/SAE, the COM/CRA, or trained site personnel will follow Section 13 of this protocol. If the AE/SAE was potentially the result of a product quality related deficiency, these procedures also applies and will be executed in parallel.

In some cases, a PQC form may be generated in EDC by the site in error. In this event, the PQC forms will be marked "Intentionally Left Blank" or "ILB". Justification for ILB must be documented.

#### 13. ADVERSE EVENTS

#### 13.1. Definitions and Classifications

**Adverse Event (AE)** – An AE is "any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users or other persons, whether or not related to the investigational medical device. This definition includes events related to the investigational medical device or the comparator, and to the procedures involved. For users or other persons, this definition is restricted to events related to investigational medical devices<sup>1</sup>

An AE includes any condition (including a pre-existing condition) that:

- 1. Was not present prior to the study, but appeared or reappeared following initiation of the study.
- 2. Was present prior to the study, but worsened during the study. This would include any condition resulting from concomitant illnesses, reactions to concomitant medications, or progression of disease states.
- 3. Pregnancy must be documented as an adverse event and must be reported to the clinical monitor and to the Sponsor immediately upon learning of the event.

Serious Adverse Event (SAE) – An SAE is any adverse event that led to any of the following:

- Death
- Serious deterioration in the health of the subject that resulted in any of the following:
- Life-threatening illness or injury
- Permanent or persistent impairment of a body structure or a body function
- Hospitalization or prolongation of patient hospitalization
- Medical or surgical intervention to prevent life-threatening illness or injury or permanent impairment to a body structure or a body function.
- Chronic disease
- Fetal distress, fetal death or a congenital physical or mental impairment of birth defect.

Diagnoses and conditions that are considered Ocular Serious Adverse Events include, but not limited to:

- Microbial Keratitis (MK)
- Iritis (including cells in the anterior chamber)
- Permanent decrease in best spectacle corrected visual acuity equivalent to 2 acuity lines or greater
- Central Corneal Opacity
- Central Corneal Neovascularization
- Uveitis
- Endophthalmitis
- Hypopyon
- Hyphemia
- Penetration of Bowman's Membrane
- Persistent Epithelial Defect

• Limbal cell Damage leading to Conjunctivalization

**Significant Adverse Events** – are defined as events that are symptomatic and warrant discontinuation (temporary or permanent) of the contact lens wear

Diagnoses and conditions that are considered Ocular Significant Adverse Events include, but not limited to the following:

- Contact Lens Induced Peripheral Ulcer (CLPU)
- Significant Infiltrative Events (SIE)
- Superior Epithelial Arcuate Lesions (SEALs)
- Any Temporary Loss of > 2 Lines of BSCVA
- Other grade 3 or higher corneal findings, such as abrasions or edema
- Non-contact lens related corneal events e.g. Epidemic Keratoconjunctivitis (EKC)
- Asymptomatic Corneal Scar
- Any corneal event which necessitates temporary lens discontinuation > 2 weeks

**Non-Significant Adverse Events** – are defined as those events that are usually asymptomatic and usually do not warrant discontinuation of contact lens wear but may cause a reduction in wear time. However, the Investigator may choose to prescribe treatment as a precautionary measure.

Diagnoses and conditions that are considered Ocular Non-Significant Adverse Events include, but not limited to the following:

- Non-significant Infiltrative Event (NSIE)
- Contact Lens Papillary Conjunctivitis (CLPC)
- Superficial Punctate Keratitis (SPK)
- Conjunctivitis: Bacterial, Viral, Allergic
- Blepharitis
- Meibomianitis
- Contact Dermatitis
- Localized Allergic Reactions
- Any corneal event not explicitly defined as serious or significant adverse event, which necessitates temporary lens discontinuation < 2 weeks

**Adverse Device Effect (ADE)** – An ADE is an "adverse event related to the use of an investigational medical device.

**NOTE 1:** to entry: This definition includes adverse events resulting from insufficient or inadequate instructions for use, deployment, implantation, installation, or operation, or any malfunction of the investigational medical device.

**NOTE 2** to entry: This definition includes any event resulting from use error or from intentional misuse of the investigational medical device."<sup>1</sup>

Unanticipated Adverse Device Effect (UADE) – Any serious adverse effect on health or safety or any life-threatening problem or death caused by, or associated with, the test article,

if that effect, problem, or death was not previously identified in nature, severity, or degree of incidence in the investigational plan, Investigator's Brochure or protocol, or any other unanticipated serious problem associated with the test article that relates to the rights, safety and welfare of subjects.

## 13.2. Assessing Adverse Events

In conjunction with the medical monitor, the Investigator will evaluate adverse events to ensure the events are categorized correctly. Elements of categorization will include:

- Seriousness/Classifications (see definition in Section 13.1).
- Causality or Relatedness i.e. the relationship between the test article, study treatment or study procedures and the adverse event (not related; unlikely related; possibly related; related see definition in Section 13.2.1).
- Adverse Event Severity Adverse event severity is used to assess the degree of intensity of the adverse event (mild; moderate; severe for all events see definition in Section 0).
- Outcome not recovered or not resolved; recovering or resolving; recovered or resolved with sequelae; recovered or resolved; death related to adverse event; unknown.
- Actions Taken none; temporarily discontinued; permanently discontinued; other.

## 13.2.1. Causality Assessment

Causality Assessment – A determination of the relationship between an adverse event and the test article. The test article relationship for each adverse event should be determined by the investigator using these explanations:

- Not Related- An adverse event that is not related to the use of the test article, study treatment or study procedures.
- Unlikely Related An adverse event for which an alternative explanation is more likely, e.g. concomitant treatment, concomitant disease(s), or the relationship of time suggests that a causal relationship is not likely.
- Possibly Related An adverse event that might be due to the use of the test article, or to the study treatment or study procedures. An alternative explanation, e.g. concomitant treatment, concomitant disease(s), is inconclusive. The relationship in time is reasonable. Therefore, the causal relationship cannot be excluded.
- Related An adverse event that is listed as a possible adverse effect (device) or adverse reaction (drug) and cannot be reasonably explained by an alternative explanation, e.g. concomitant treatment of concomitant disease(s). The relationship in time is very suggestive, e.g. it is confirmed by de-challenge and re-challenge.

#### 13.2.2. Severity Assessment

**Severity Assessment** – A qualitative assessment of the degree of intensity of an adverse event as determined by the Investigator or reported to him/her by the subject. The assessment of severity is made irrespective of test article, study treatment or study procedure relationship or seriousness of the event and should be evaluated according to the following scale:

- Mild Event is noticeable to the subject, but is easily tolerated and does not interfere with the subject's daily activities.
- Moderate Event is bothersome, possible requiring additional therapy, and may interfere with the subject's daily activities.
- Severe Event is intolerable, necessitates additional therapy or alteration of therapy and interferes with the subject's daily activities.

## 13.3. Documentation and Follow-Up of Adverse Events

The recording and documenting of adverse events (ocular and non-ocular) begin when the subjects are exposed to the test article, study treatment or study procedure. Adverse events reported before the use of test article, start of study treatment, or study procedures will be recorded as medical history. However, if the condition deteriorates at any time during the study it will be recorded and reported as an AE. Untoward medical events reported after the subject's exit from the study will be recorded as adverse events at the discretion of the Investigator.

Upon finding an adverse event, the Principal Investigator will document the condition in the subject record and in the eCRFs. He/she will complete the Adverse Event /eCRF.

Complete descriptions of all adverse events must be available in the subject record. All Adverse Events including local and systemic reactions not meeting the criteria for "serious adverse events" shall be captured on the appropriate case report form or electronic data system. All adverse events occurring while the subject is enrolled in the study must be documented appropriately regardless of relationship.

It is the Investigator's responsibility to maintain documentation of each reported adverse event. All adverse events will be followed in accordance with applicable licensing requirements. Such documentation will include the following:

- Adverse event (diagnosis not symptom).
- Drawings or photographs (where appropriate) that detail the finding (e.g., size, location, and depth, etc.).
- Date the clinical site was notified.
- Date and time of onset.
- Date and time of resolution.
- Adverse event classification, severity, and relationship to test articles, as applicable.
- Treatment regimen instituted, including concomitant medications prescribed, in accordance with applicable licensing requirements.
- Any referral to another health care provider if needed.
- Outcome, ocular damage (if any).
- Likely etiology.
- Best corrected visual acuity at the discovery of the event and upon conclusion of the event, if related to the visual system.

In addition, if an infiltrate(s) is present, he/she will complete the Corneal Infiltrate Assessment eCRF. Where necessary, a culture of the corneal lesion will be collected to determine if the

infection is microbial in nature. If cultures are collected, the date of culture collection and laboratory utilized will be recorded.

Changes in the severity of an AE shall be documented to allow an assessment of the duration of the event at each level of intensity to be performed. Adverse events characterized as intermittent require documentation of the onset and duration of each episode. Changes in the assessment of relationship to the Test Article shall also be clearly documented.

Subjects who present with an adverse event shall be followed by the Investigator, within licensure, until all signs and symptoms have returned to pre-treatment status, stabilized, or been satisfactorily resolved. If further treatment beyond licensure is required, the patient will be referred to the appropriate health care provider. The Investigator will use his/her clinical judgment as to whether a subject reporting with an adverse event will continue in the study. If a subject is discontinued from the study, it will be the responsibility of the Investigator to record the reason for discontinuation. The Investigator will also document the adverse event appropriately and complete the Adverse Event eCRF. Any subjects with ongoing adverse events related to the test article, study treatment or study procedures, as of the final study visit date, should be followed to resolution of the adverse event or until referral to an appropriate health care provider, as recommended by the Investigator. Non-ocular adverse events that are not related to the test article, study treatment, or study procedures may be recorded as "ongoing" without further follow-up.

## 13.4. Reporting Adverse Events

The Investigator will notify the Sponsor of an adverse event by e-mail, facsimile, or telephone as soon as possible and no later than 24 hours from discovery for any serious /significant adverse events, and 2 days from discovery for any non-significant adverse event. In addition, a written report will be submitted by the Principal Investigator to the IEC/IRB according to their requirements (Section 13.4.2). The report will comment whether the adverse event was considered to be related to the test article, study treatment or study procedures.

#### 13.4.1. Reporting Adverse Events to Sponsor

## **Serious/Significant Adverse Events**

The Investigator will inform the sponsor of all serious/significant adverse events occurring during the study period as soon as possible by e-mail, fax, or telephone, but no later than 24 hours following discovery of the event. The Investigator is obligated to pursue and obtain information requested by the Sponsor in addition to that information reported on the eCRF. All subjects experiencing a serious/significant adverse event must be followed up and all outcomes must be reported.

When medically necessary, the Investigator may break the randomization code to determine the identity of the treatment that the subject received. The Sponsor and study monitor should be notified prior to unmasking the test articles.

In the event of a serious/significant adverse event, the Investigator must:

• Notify the Sponsor immediately.

- Obtain and maintain in the subject's records all pertinent medical information and medical judgment for colleagues who assisted in the treatment and follow-up of the subject.
- Provide the Sponsor with a complete case history which includes a statement as to whether the event was or was not related to the use of the test article.
- Notify the IEC/IRB as required by the IEC/IRB reporting procedure according to national regulations.

## **Unanticipated (Serious) Adverse Device Effect (UADE)**

In the event of an Unanticipated (Serious) Adverse Device Effect (UADE), the Investigator will submit a report of the UADE to the Sponsor and IEC/IRB as soon as possible, but no later than 24 hours after the Investigator first learns of the effect. This report is in addition to the immediate notification mentioned above.

The Sponsor must conduct an evaluation of the UADE and must report the results of the evaluation to FDA, the IEC/IRB and participating Investigators within 10 working days after the Sponsor first receives notification of the effect.

#### **Non-Serious Adverse Events**

All non-serious adverse events, including non-serious adverse device effects, will be reported to the sponsor by the Investigator no later than 2 days from discovery.

## 13.4.2. Reporting Adverse Events to the Responsible IEC/IRB and Health Authorities

Adverse events that meet the IEC/IRB requirements for reporting must be reported within the IEC/IRB's written guidelines. Each clinical site will refer to and follow any guidelines set forth by their Approving IEC/IRB. Each clinical site will refer to and follow any guidelines set forth by their local governing Health Authorities.

The Sponsor will report applicable Adverse Events to the local health authorities according the written guidelines, including reporting timelines.

## 13.4.3. Event of Special Interest

Not applicable

#### 13.5. Reporting of Pregnancy

Subjects reporting pregnancy (by self-report) during the study will be discontinued after the event is recorded as an Adverse Event. Once discontinued, pregnant participants and their fetuses will not be monitored for study related purposes. At the Investigator's discretion, the study participant may be followed by the Investigator through delivery. However, this data will not be collected as part of the clinical study database. Pregnant participants are not discontinued from contact lens or solution related studies for safety concerns, but due to general concerns relating to pregnancy and contact lens use. Specifically, pregnant women are discontinued due to fluctuations in refractive error and/or visual acuity that occur secondary to systemic hormonal changes, and not due to unforeseen health risks to the mother or fetus.

#### 14. STATISTICAL METHODS

## 14.1. General Considerations

Statistical analysis will be undertaken by the study biostatistician. A general description of the statistical methods to be implemented in this clinical trial is outlined below.

All data summaries and statistical analyses will be performed using the SAS software Version 9.4 or higher (SAS Institute, Cary, NC). Throughout the analysis of data, the results for each subject/eye will be used when available for summarization and statistical analysis.

Summary tables (descriptive statistics and/or frequency tables) will be provided for all baseline variables, efficacy variables, and safety variables as appropriate. Continuous variables will be summarized with descriptive statistics (n, mean, standard deviation [SD], median, minimum and maximum). Frequency count and percentage of subjects or eyes within each category will be provided for categorical data.

## 14.2. Sample Size Justification

This study was not designed or powered to test any statistical hypotheses. The purpose of this study is to assess the performance of the study lenses with respect to distance and near visual acuity (logMAR), qCSF and qVA. Therefore, the sample size of 30 subjects to enroll with approximately 25 subjects to complete the study will be sufficient to evaluate the performance of the study lenses with respect to the primary endpoint.

## 14.3. Analysis Populations

## **Safety Population:**

All subjects who were administered any test article excluding subjects who drop out prior to administering any test article. At least one observation should be recorded.

#### **Per-Protocol Population:**

All subjects who have successfully completed all visits and did not substantially deviate from the protocol as determined by the trial cohort review committee prior to database hard lock (Per-Protocol Population). Justification of excluding subjects with protocol deviations in the Per-Protocol Population set will be documented in a memo to file.

## **Intent-to-Treat (ITT) Population:**

All randomized subjects regardless of actual treatment and subsequent withdrawal from study or deviation from protocol. At least one observation should be recorded.

#### 14.4. Level of Statistical Significance

Not applicable

## 14.5. Primary Analysis

Distance and near visual acuity, qCSF and qVA will be descriptively summarized by lens type.

## 14.6. Secondary Analysis

Not applicable.

## 14.7. Other Exploratory Analyses

Further statistical exploratory analysis can be undertaken, if necessary, at the discretion of the clinical project leader.

## 14.8. Interim Analysis

An interim analysis will not be conducted on this study.

# 14.9. Procedure for Handling Missing Data and Drop-Outs

Missing or spurious values will not be imputed. The count of missing values will be included in the summary tables and listings.

## 14.10. Procedure for Reporting Deviations from Statistical Plan

The analysis will be conducted according to that specified in above sections. There are no known reasons for which it is planned to deviate from these analysis methods. If for any reason a change is made, the change will be documented in the study report along with a justification for the change.

#### 15. DATA HANDLING AND RECORD KEEPING/ARCHIVING

#### 15.1. Electronic Case Report Form/Data Collection

The data for this study will be captured on electronic case report forms (eCRFs) using an EDC system (Bioclinica Express 5.5). An authorized data originator will enter study data into the eCRFs using the EDC system. Data collected on equipment that is not captured in EDC will be formatted to the specification of the JJVC database manager and sent to JJVC for analysis.

External Data Sources for this study include: Not Applicable

The clinical data will be recorded on dedicated eCRFs specifically designed to match the study procedures for each visit. Only specifically delegated staff can enter data on a CRF. Once completed, the eCRFs will be reviewed for accuracy and completeness and signed by the Investigator. The sponsor or sponsor's representatives will be authorized to gain access to the subject recordation for the purposes of monitoring and auditing the study.

Edit checks, electronic queries, and audit trails are built into the system to ensure accurate and complete data collection. Data will be transmitted from the clinical site to a secure central database as forms are completed or updated, ensuring information accuracy, security, and confidentiality. After the final database lock, the Investigator will be provided with Individual Patient Profiles (IPP) including the full audit trail on electronic media in PDF format for all of the study data. The IPP must be retained in the study files as a certified copy of the source data for the study.

The content and structure of the eCRFs are compliant with ISO14155:2011.<sup>1</sup>

## 15.2. Subject Record

At a minimum, subject record should be available for the following:

- subject identification
- eligibility
- study identification
- study discussion
- provision of and date of informed consent
- visit dates
- results of safety and efficacy parameters as required by the protocol
- a record of all adverse events
- follow-up of adverse events
- medical history and concomitant medication
- test article receipt/dispensing/return records
- date of study completion
- reason for early discontinuation of test article or withdrawal from the study, if applicable

The subject record is the eCRF or an external record. The author of an entry in the subject record must be identifiable. The first point of entry is considered to be the source record.

Adverse event notes must be reviewed and initialed by the Investigator.

#### 15.3 ClinicalTrials.gov

This study will be registered on ClinicalTrials.gov based on the following: confirmatory study meets the requirements for registration.

#### 16. DATA MANAGEMENT

#### 16.1. Access to Source Data/Document

The Investigator/Institution will permit trial-related monitoring, audits, IEC/IRB review and regulatory inspection(s) by providing direct access to source data/documents. Should the clinical site be contacted for an audit by an IEC/IRB or regulatory authority, JJVC must be contacted and notified in writing within 24 hours.

## 16.2. Confidentiality of Information

Information concerning the investigational product and patent application processes, scientific data or other pertinent information is confidential and remains the property of JJVC. The Investigator may use this information for the purposes of the study only. It is understood by the Investigator that JJVC will use information developed in this clinical study in connection

with the development of the investigational product and therefore may disclose it as required to other clinical investigators and to regulatory agencies. In order to allow the use of the information derived from this clinical study, the Investigator understands that he/she has an obligation to provide complete test results and all data developed during this study to the Sponsor.

## 16.3. Data Quality Assurance

Steps will be taken to ensure the accuracy and reliability of data, include the selection of qualified investigators and appropriate clinical sites and review of protocol procedures with the Principal Investigator. The Principal Investigator, in turn, must ensure that all Sub-Investigators and clinical site personnel are familiar with the protocol and all study-specific procedures and have appropriate knowledge of the study article.

Training on case report form completion will be provided to clinical site personnel before the start of the study. The Sponsor will review case report forms for accuracy and completeness remotely during the conduct of the study, during monitoring visits, and after transmission to data management. Any data discrepancies will be resolved with the Investigator or designee, as appropriate.

Quality Assurance representatives from JJVC may visit clinical sites to review data produced during the study and to access compliance with applicable regulations pertaining to the conduct of clinical trials. The clinical sites will provide direct access to study-related source data/documents and reports for the purpose of monitoring and auditing by JJVC and for inspection by local and regulatory authorities.

## 17. CLINICAL MONITORING

The study monitors will maintain close contact with the Principal Investigator and the Investigator's designated clinical site personnel. The monitor's responsibilities will include:

- Ensuring that the investigation is being conducted according to the protocol, any subsequent versions, and regulatory requirements are maintained.
- Ensuring the rights and wellbeing of subjects are protected.
- Ensuring adequate resources, including facilities, laboratories, equipment, and qualified clinical site personnel.
- Ensuring that protocol deviations are documented with corrective action plans, as applicable.
- Ensuring that the clinical site has sufficient test article and supplies.
- Clarifying questions regarding the study.
- Resolving study issues or problems that may arise.
- Reviewing of study records and source documentation verification in accordance with the monitoring plan.

#### 18. ETHICAL AND REGULATORY ASPECTS

## 18.1. Study-Specific Design Considerations

Potential subjects will be fully informed of the risks and requirements of the study and, during the study, subjects will be given any new information that may affect their decision to continue participation. Subjects will be told that their consent to participate in the study is voluntary and may be withdrawn at any time with no reason given and without penalty or loss of benefits to which they would otherwise be entitled. Only subjects who are fully able to understand the risks, benefits, and potential adverse events of the study, and provide their consent voluntarily will be enrolled.

## 18.2. Investigator Responsibility

The Principal Investigator is responsible for ensuring that the clinical study is performed in accordance with the signed agreement, the investigational plan, Section 4 of the ICH E6 guidelines on Good Clinical Practice (GCP),<sup>2</sup> and applicable regulatory requirements. GCP is an international ethical and scientific quality standard for designing, conducting, recording, and reporting studies that involve the participation of human subjects. Compliance with this standard provides public assurance that the rights, safety, and well-being of study subjects are protected, consistent with the principles of the Declaration of Helsinki 64<sup>th</sup> WMA General Assembly 2013<sup>3</sup> and that the clinical study data are credible. The Investigator must maintain clinical study files in accordance with Section 8 of the ICH E6 guidelines on Good Clinical Practice (GCP),<sup>2</sup> and applicable regulatory requirements.

## 18.3. Independent Ethics Committee or Institutional Review Board (IEC/IRB)

Before the start of the study, the Investigator (or Sponsor when applicable) will provide the IEC/IRB with current and complete copies of the following documents (where applicable):

- Final protocol.
- Sponsor-approved informed consent form (and any other written materials to be provided to the subjects)
- Investigator's Brochure (or equivalent information).
- Sponsor-approved subject recruitment materials.
- Information on compensation for study-related injuries or payment to subjects for participation in the study.
- Investigator's curriculum vitae, clinical licenses, or equivalent information (unless not required, as documented by IEC/IRB).
- Information regarding funding, name of the Sponsor, institutional affiliations, other potential conflicts of interest, and incentives for subjects.
- Any other documents that the IEC/IRB requests to fulfill its obligation.

This study will be undertaken only after IEC/IRB has given full approval of the final protocol, the informed consent form, applicable recruiting materials, and subject compensation programs, and the Sponsor has received a copy of this approval. This approval letter must be dated and must clearly identify the documents being approved.

During the study, the Investigator (or Sponsor when applicable) will send the following documents to the IEC/IRB for their review and approval, where appropriate:

- Protocol revisions
- Revision(s) to informed consent form and any other written materials to be provided to subjects
- If applicable, new or revised subject recruitment materials approved by the Sponsor
- Revisions to compensation for study-related injuries or payment to subjects for participation in the study
- Investigator's Brochure revisions
- Summaries of the status of the study (at least annually or at intervals stipulated in guidelines of the IEC/IRB)
- Reports of adverse events that are serious, unanticipated, and associated with the test articles, according to the IRB's requirements
- New information that may adversely affect the safety of the subjects or the conduct of the study
- Major protocol deviations as required by the IEC/IRB
- Report of deaths of subjects under the Investigator's care
- Notification if a new Investigator is responsible for the study at the clinical site
- Any other requirements of the IEC/IRB

For protocol revisions that increase subject risk, the revisions and applicable informed consent form revisions must be submitted promptly to the IEC/IRB for review and approval before implementation of the change(s).

At least once a year, the IEC/IRB will review and reapprove this clinical study. This request should be documented in writing.

At the end of the study, the Investigator (or Sponsor where required) will notify the IEC/IRB about the study completion. Documentation of this notification must be retained at the clinical site and a copy provided to the CRO or Sponsor as applicable.

#### 18.4. Informed Consent

Each subject or their representative, must give written consent according to local requirements after the nature of the study has been fully explained. The consent form must be signed before performance of any study-related activity. The consent form that is used must be approved by both the Sponsor and by the reviewing IEC/IRB. The informed consent is in accordance with principles that originated in the Declaration of Helsinki,<sup>3</sup> current ICH<sup>2</sup> and ISO 14155<sup>1</sup> guidelines, applicable regulatory requirements, and Sponsor Policy.

Before entry into the study, the Investigator or an authorized member of the clinical site personnel must explain to potential subject the aims, methods, reasonably anticipated benefits, and potential hazards of the study, and any discomfort it may entail. Subjects will be informed that their participation is voluntary and that they may withdraw consent to participate at any time.

The subject will be given sufficient time to read the informed consent form and the opportunity to ask questions. After this explanation and before entry into the study, consent should be appropriately recorded by means of the subject's dated signature. After having obtained the consent, a copy of the informed consent form must be given to the subject.

Each subject for this study will complete an assent and a parent or legal guardian must give written informed consent according to local requirements after the nature of the study has been fully explained. The assent and consent forms must be signed before performance of any studyrelated activity. The assent and consent forms that are used must be approved by both the Sponsor and by the reviewing IEC/IRB. The assent and informed consent forms should be in accordance with principles that originated in the Declaration of Helsinki,<sup>3</sup> current ICH<sup>2</sup> and GCP guidelines, applicable regulatory requirements, and Sponsor policy. Before entry into the study or pre-screening, the Investigator or an authorized member of the clinical site personnel must explain to the potential subject and parent and/or legal guardian the aims, methods, reasonably anticipated benefits, and potential hazards of the study or pre-screening, and any discomfort it may entail. Subjects and parent and/or legal guardian will be informed that their participation is voluntary and that they may withdraw consent to participate at any time. They will be informed that choosing not to participate will not affect the care the subject will receive. Finally, they will be told that the Investigator will maintain a subject identification register for the purposes of long-term follow-up if needed and that their records may be accessed by health authorities and authorized Sponsor personnel without violating the confidentiality of the subject, to the extent permitted by the applicable law(s) or regulations. By signing the assent and informed consent form, the subject is authorizing such access and agrees to be contacted after study completion by health authorities and authorized Sponsor personnel for the purpose of obtaining consent for additional safety evaluations if needed.

#### 18.5. Privacy of Personal Data

The collection, processing and disclosure of personal data and medical information related to the Study Subject, and personal data related to Principal Investigator and any clinical site personnel (e.g., name, clinic address and phone number, curriculum vitae) is subject to compliance with the Health Information Portability and Accountability Act (HIPAA) in the United States<sup>7</sup> and other applicable personal data protection and security laws and regulations. Appropriate measures will be employed to safeguard these data, to maintain the confidentiality of the person's related health and medical information, to properly inform the concerned persons about the collection and processing of their personal data, to grant them reasonable access to their personal data and to prevent access by unauthorized persons.

All information obtained during the course of the investigation will be regarded as confidential. All personal data gathered in this trial will be treated in strictest confidence by Investigators, monitors, Sponsor's personnel and IEC/IRB. No data will be disclosed to any third party without the express permission of the subject concerned, with the exception of Sponsor personnel (monitor, auditor), IEC/IRB and regulatory organizations in the context of their investigation related activities that, as part of the investigation will have access to the CRFs and subject records.

The collection and processing of personal data from subjects enrolled in this study will be limited to those data that are necessary to investigate the efficacy, safety, quality, and utility of the investigational product(s) used in this study.

These data must be collected and processed with adequate precautions to ensure confidentiality and compliance with applicable data privacy protection laws and regulations.

The Sponsor ensures that the personal data will be:

- processed fairly and lawfully.
- collected for specified, explicit, and legitimate purposes and not further processed in a way incompatible with these purposes.
- adequate, relevant, and not excessive in relation to said purposes.
- accurate and, where necessary, kept current.

Explicit consent for the processing of personal data will be obtained from the participating subject before collection of data. Such consent should also address the transfer of the data to other entities and to other countries.

The subject has the right to request through the Investigator access to his personal data and the right to request rectification of any data that are not correct or complete. Reasonable steps should be taken to respond to such a request, taking into consideration the nature of the request, the conditions of the study, and the applicable laws and regulations.

Appropriate technical and organizational measures to protect the personal data against unauthorized disclosures or access, accidental or unlawful destruction, or accidental loss or alteration must be put in place. Sponsor personnel whose responsibilities require access to personal data agree to keep the identity of study subjects confidential.

#### 19. STUDY RECORD RETENTION

In compliance with the ICH/GCP guidelines,<sup>2</sup> the Investigator/Institution will maintain all CRFs and all subject records that support the data collected from each subject, as well as all study documents as specified in ICH/GCP<sup>2</sup> and all study documents as specified by the applicable regulatory requirement(s). The Investigator/Institution will take measures to prevent accidental or premature destruction of these documents.

Essential documents must be retained until at least two (2) years after the last approval of a marketing application in an ICH region and until there are no pending or contemplated marketing applications in an ICH region or until at least two (2) years have elapsed since the formal discontinuation of clinical development of the investigational product. These documents will be retained for a longer period if required by the applicable regulatory requirements or instructed by the Sponsor. It is the responsibility of the Sponsor to inform the Investigator/Institution as to when these documents no longer need to be retained.

If the responsible Investigator retires, relocates, or for other reasons withdraws from the responsibility of keeping the study records, custody must be transferred to a person who will

accept the responsibility. The Sponsor must be notified in writing of the name and address of the new custodian. Under no circumstance shall the Investigator relocate or dispose of any study documents before having obtained written approval from the Sponsor.

If it becomes necessary for the Sponsor or the appropriate regulatory authority to review any documentation relating to this study, the Investigator must permit access to such reports. If the Investigator has a question regarding retention of study records, he/she should contact JJVC.

#### 20. FINANCIAL CONSIDERATIONS

Remuneration for study services and expenses will be set forth in detail in the Clinical Research Agreement. The Research Agreement will be signed by the Principal Investigator and a JJVC management representative prior to study initiation.

JJVC reserves the right to withhold remuneration for costs associated with protocol violations such as:

- Continuing an ineligible subject in the study.
- Scheduling a study visit outside the subject's acceptable visit range.

JJVC reserves the right to withhold final remuneration until all study related activities have been completed, such as:

- Query resolution.
- Case Report Form signature.
- Completion of any follow-up action items.

#### 21. PUBLICATION

This study will be registered on ClinicalTrials.gov by the Sponsor.

#### 22. REFERENCES

- 1. ISO 14155:2011: Clinical Investigation of Medical Devices for Human Subjects Good Clinical Practice. Available at: https://www.iso.org/standard/45557.html
- 2. International Conference on Harmonization Good Clinical Practice E6 (ICH-GCP). Available at: http://www.ich.org/products/guidelines/efficacy/article/efficacy-guidelines.html
- 3. Declaration of Helsinki Ethical principles for Medical Research Involving Human Subjects. Available at: https://www.wma.net/policies-post/wma-declaration-of-helsinki-ethical-principles-for-medical-research-involving-human-subjects/
- 4. United States (US) Code of Federal Regulations (CFR). Available at: https://www.gpo.gov/fdsys/browse/collectionCfr.action?collectionCode=CFR
- 5. Wirth RJ, et al. Development of the Contact Lens User Experience: CLUE Scales. *Optom Vis Sci.* 2016;93(8):801-808

6.

- 7. Health Information Portability and Accountability Act (HIPAA). Available at: https://www.hhs.gov/hipaa/for-professionals/privacy/index.html
- 8. EU MDR 2017/745

APPENDIX A: PATIENT REPORTED OUTCOMES (STUDY QUESTIONNAIRES)












# APPENDIX B: PATIENT INSTRUCTION GUIDE

This will be provided separately.

APPENDIX C: PACKAGE INSERT (APPROVED PRODUCT)

1-DAY ACUVUE® DEFINE™ Brand Contact Lenses

| Example 1 | |
|----------------------------|--------|
| Diagnostic lens: | -2.00D |
| Spherical over-refraction: | -0.25D |
| Final lens power: | -2.25D |

| Example 2 | |
|----------------------------|--------|
| Diagnostic lens: | -2.00D |
| Spherical over-refraction: | +0.25D |
| Final lens power: | -1.75D |

If vision is acceptable, perform a slit lamp examination to confirm adequate fit (centration and movement), if the fit is acceptable, dispense the lenses and instruct the patient to return in one week for reassessment (see dispensing and follow up information in PATIENT MANAGEMENT).

All patients should be supplied with a copy of the "1-DAY ACUVUE® DEFINE™ Brand Contact Lenses Patient Instruction Guide." Copies are available for download at www.acuvue.com.

#### MONOVISION FITTING GUIDELINES

#### A. Patient Selection

#### Monovision Needs Assessment

For a good prognosis, the patient should have adequately corrected distance and near visual acuity in each eye. The amblyopic patient with significant astigmatism (greater than 1.00D) in one eye may not be a good candidate for monovision correction with the 1-DAY ACUVUE® DEFINE® Contact Lenses.

Occupational and environmental visual demands should be considered. If the patient requires critical vision (visual acuity and stereopsis), it should be determined by trial whether this patient can function adequately with monovision correction. Monovision contact lens wear may not be optimal for such activities as:

- visually demanding situations such as operating potentially dangerous machinery or performing other potentially hazardous activities; and
- 2.driving automobiles (e.g., driving at night). Patients who cannot pass their state driver's license

#### Every three to six months thereafter

NOTE: Preferably, at the follow-up visits, lenses should be worn for at least six hours.

#### B. Recommended Procedures for Follow-Up Visits:

- 1. Solicit and record patient's symptoms, if any.
- Measure visual aculty monocularly and binocularly at distance and near with the contact lenses.
- Perform an over-refraction at distance and near to check for residual refractive error.
- With the biomicroscope, judge the lens fitting characteristics (as described in the GENER-AL FITTING GUIDELINES) and evaluate the lens surface for deposits and damage.
- Following lens removal, examine the cornea and conjunctiva with the biomicroscope and fluorescein (unless contraindicated).
  - The presence of vertical corneal striae in the posterior central cornea and/or corneal neovascularization is indicative of excessive corneal edema.
  - The presence of corneal staining and/or limbal-conjunctival hyperemia can be indicative of an unclean lens, a reaction to solution preservatives, excessive lens wear and/or a poorly fitting lens.
- Papillary conjunctival changes may be indicative of an unclean and/or damaged lens.

  Postediculty perform terretometry and executed performance. The values obserted by reported.
- Periodically perform keratometry and spectacle refractions. The values should be recorded and compared to the baseline measurements.

If any observations are abnormal, use professional judgment to alleviate the problem and restore the eye to optimal conditions. If the criteria for successful fit are not satisfied during any follow-up examinations, repeat the patient's trial fitting procedure and refit the patient.

#### WEARING SCHEDULE

The wearing schedule should be determined by the Eye Care Professional. Regular checkups, as determined by the Eye Care Professional, are also extremely important.

Patients tend to over wear the lenses initially. The Eye Care Professional should emphasize the importance of adhering to the initial maximum wearing schedule. Maximum wearing time should be determined by the Eye Care Professional based upon the patient's physiological eye condition, because individual response to contact lenses varies.

CR-6396, v 2.0

requirements with monovision correction should be advised to not drive with this correction, or may require that additional over-correction be prescribed.

#### Patient Education

All patients do not function equally well with monovision correction. Patients may not perform as well for certain tasks with this correction as they have with spectacles (multifocal, bifocal, trifocal, readers or progressives). Each patient should understand that monovision, as well as other presbyopic alternatives, can create a vision compromise that may reduce visual acuity and depth perception for distance and near tasks. Therefore, caution should be exercised. During the fitting process, it is necessary for the patient to realize the disadvantages as well as the advantages of clear near vision and straight ahead and upward gaze that monovision contact lenses provide.

#### B. Eye Selection

Generally, the non-dominant eye is corrected for near vision. The following two methods for eye dominance can be used.

#### 1. Ocular Preference Determination Methods

Method 1: Determine which eye is the "sightling eye." Have the patient point to an object at the far end of the room. Cover one eye. If the patient is still pointing directly at the object, the eye being used is the dominant (sightling) eye.

Method 2: Determine which eye will accept the added power with the least reduction in vision. Place a hand-held trial lens equal to the spectacle near ADD in front of one eye and then the other while the distance refractive error correction is in place for both eyes. Determine whether the patient functions best with the near ADD lens over the right or left eye.

Other methods include the "Refractive Error Method" and the "Visual Demands Method."

#### 2. Refractive Error Method

For anisometropic correction, it is generally best to fit the more hyperopic (less myopic) eye for distance and the more myopic (less hyperopic) eye for near.

#### 3 Vieual Demande Method

Consider the patient's occupation during the eye selection process to determine the critical vision requirements. If a patient's gaze for near tasks is usually in one direction, correct the eve on that side for near.

The maximum suggested wearing time for these lenses is:

| DAYS | HOURS |
|-------------|------------------|
| 1 | 6-8 |
| 2 | 8-10 |
| 3 | 10-12 |
| 4 | 12-14 |
| 5 and after | all waking hours |

#### REPLACEMENT SCHEDULE

1-DAY ACUVUE® DEFINE™ Contact Lenses when prescribed for daily disposable wear should be discarded upon removal.

When disposed of after a single daily use, these lenses may reduce the risk of developing giant papillary conjunctivitis.<sup>4</sup>

When worn as a daily disposable lens, the lenses may provide improved comfort for many patients who experience mild discomfort and litching associated with allergies during contact lens wear, compared to lenses replaced at intervals of greater than 2 weeks.

Clinical Research has shown that when worn on a daily disposable basis, these lenses may provide improved comfort for 2 out of 3 patients who reported suffering from discomfort associated with allergies during contact lens wear.

<sup>4</sup>The CLAO Journal, July 1999, Volume 25, Number 3

#### LENS CARE DIRECTIONS

When lenses are prescribed for daily disposable wear, the Eye Care Professional should provide the patient with appropriate and adequate warnings and instructions for daily disposable lens wear at the time they are dispensed.

The Eye Care Professional should review with patients that no cleaning or disinfection is needed with daily disposable lenses. Patients should always dispose of lenses when they are removed and have spare lenses or spectacles available.

#### Basic Instructions

- Always wash, rinse, and dry hands before handling contact lenses.
- Do not use saliva or anything other than the recommended solutions for lubricating or rewetting lenses. Do not put lenses in the mouth.

Example: A secretary who places copy to the left side of the desk will near lens on the left eye.

#### C. Special Fitting Characteristics

#### 1. Unilateral Vision Correction Requirement

There are circumstances where only one contact lens is require tion purposes (e.g., presbyopic emmetripoc patient would only whereas a bilateral myope would require corrective lenses on b

Due to the indication of altering and/or enhancing the natural a eye, the non-corrected eye may be fit with a 0.00D lens to ens

Example: A presbyopic emmetropic patient who requires a +1.75D ADD wor on the near eye and a 0.00D lens (uncorrected) may be fit on the other eye.

A presbyopic patient requiring a +1.500 ADD who is -2.500 myopic in the myopic in the left eye may have the right eye corrected for distance and the a 0.000 lens (uncorrected) for near.

#### 2. Near ADD Determination

Always prescribe the lens power for the near eye that provides at the midpoint of the patient's habitual reading distance. How than one power provides optimal reading performance, prescri (most minus) of the powers.

#### 3. Trial Lens Fitting

A trial fitting is performed in the office to allow the patient to ex sion correction. Lenses are fit according to the **GENERAL FIT LINES** for base curve selection described in this guide.

Case history and standard clinical evaluation procedure should determine the prognosis. Determine the distance correction artion. Next determine the near ADD. With trial lenses of the proposerve the reaction to this mode of correction.

Allow the lenses to settle for about 20 minutes with the correct in place. Walk across the room and have the patient look at yo patient's reaction to distance vision under these circumstances patient look at familiar near objects such as a watch face or fin assess the reaction. As the patient continues to look around the near and distance objects, observe the reactions. Only after the completed should the patient be asked to read print. Evaluate

 Eye Care Professionals may recommend a lubricating/rewett can be used to wet (lubricate) lenses while they are being we more comfortable.

#### Care for a Sticking (Non-Moving) Lens

If the lens sticks (stops moving), the patient should be instructed drops of the recommended lubricating or rewetting solution dire wait until the lens begins to move freely on the eye before remov ment of the lens continues after a few minutes, the patient shoul consult the Eye Care Professional.

#### **EMERGENCIES**

The patient should be informed that if chemicals of any kind (hou gardening solutions, laboratory chemicals, etc.) are splashed into then should: FLUSH EYES IMMEDIATELY WITH TAP WATER ALL CONTACT THE EYE CARE PROFESSIONAL OR VISIT A HOSP ROOM WITHOUT DELAY.

#### **HOW SUPPLIED**

Each sterile lens is supplied in a foll-sealed plastic package cont saline solution with povidone. The plastic package is marked wit diameter, diopter power, variant, lot number, and expiration date



#### SYMBOLS KEY

The following symbols may appear on the label or carton:

| SYMBOL | DEFINITION |
|---|---|
| | Consult Instructions for Use |
| m | Date of Manufacture |
| - | Manufactured by or in |
| Z | Use By Date (expiration date) |
| LOT | Batch Code |
| DEPAG | Sterile Using Steam or Dry Heat |
| DIA | Diameter |
| BC | Base Curve |
| D | Biopter (leas power) |
| 32 | Quality System Certification Symbol |
| -F | UV-Blocking |
| 0 | Fee Paid for Waste Management |
| R <sub>Cody</sub> | CAUTION: Federal law restricts<br>this device to sale by or on the<br>order of a licensed practitioner |
| A | ACCENT STYLE |
| SH | NATURAL SHIMMERTM |
| N | NATURAL SHINE™ |
| S, | NATURAL SPARKLE™ |
| ٧ | VIVID STYLE |

#### DESCRIPTION

The 1-DAY ACUVUE® DEFINE™ Brand Contact Lenses with LACREON® Technology are soft (hydrophilic) contact lenses available as spherical lenses. The lens material (etaflicon A) is a copolymer of 2-hydroxyethyl methacrylate and methacrylic acid cross-linked with 1, 1, 1-trimethylol propane trimethacrylate and ethylene glycol dimethacrylate.

The 1-DAY ACUVUE™ DEFINE™ Brand Contact Lenses are tinted blue using Reactive Blue Dye #4 to make the lenses more visible for handling. The lenses contain a pigmented area that will after or enhance the appearance of the natural Iris. The lens is colored with one or more of the following color additives: iron oxides, titanium dioxide, phthalocyaninato (2-) copper, phythalocyanine green, and Reactive Blue Dye #4.

#### WARNING:

Water can harbor microorganisms that can lead to severe infection, vision loss or blindness. If lenses have been submersed in water when participating in water sports or swimming in pools, hot tubs, lakes or oceans, the patient should be instructed to discard them and replace them with a new pair. The Eye Care Professional should be consulted for recommendations regarding wearing lenses during any activity involving water.

#### **PRECAUTIONS**

#### Special Precautions for Eye Care Professionals:

Due to the small number of patients enrolled in clinical investigation of lenses, all refractive powers, design configurations or lens parameters available in the lens material are not evaluated in significant numbers. Consequently, when selecting an appropriate lens design and parameters, the Eye Care Professional should consider all characteristics of the lens that can affect lens performance and ocular health, including oxygen permeability, wettability, central and peripheral thickness, and cotic zone diameter.

The potential impact of these factors on the patient's ocular health should be carefully weighed against the patient's need for refractive correction; therefore, the continuing ocular health of the patient and lens performance on the eye should be carefully monitored by the prescribing Eye Care Professional.

- Patients who wear the 1-DAY ACUVUE® DEFINE™ Contact Lenses to correct presbyopia using
  monovision may not achieve the best corrected visual acuity for either far or near vision. Visual
  requirements vary with the individual and should be considered when selecting the most appropriate type of lens for each patient.
- Fluorescein, a yellow dye, should not be used while the lenses are on the eyes. The lenses
  absorb this dye and become discolored. Whenever fluorescein is used in eyes, the eyes should
  be flushed with a sterile saline solution that is recommended for in-eye use.
- Eye Care Professionals should instruct the patient to remove the lenses immediately if the eyes become red or irritated.

Eye Care Professionals should carefully instruct patients about the following care regimen and safety precautions:

#### Handling Precautions:

- Before leaving the Eye Care Professional's office, the patient should be able to promptly remove lenses or should have someone else available who can remove the lenses for him or her.
- DO NOT use if the sterile blister package is opened or damaged.
- Always wash and rinse hands before handling lenses. Do not get cosmetics, lotions, soaps,

The 1-DAY ACUVUE® DEFINE™ Contact Lenses are available in the following variants (i.e., patterns):

- ACCENT STYLE
- NATURAL SHIMMER™
- NATURAL SHINE™
- NATURAL SPARKLE™
- VIVID STYLE

A benzotriazole UV absorbing monomer is used to block UV radiation. The UV Blocking averages 97% in the UVB range of 290 nm to 315 nm and 81% in the UVA range of 316 nm to 380 nm.

#### Lens Properties:

The physical/optical properties of the lens are:

Specific Gravity (calculated): 0.98 – 1.13
 Refractive Index: 1.40
 Light Transmittance: 70% minimum
 Surface Character: Hydrophilic
 Water Content: 58%

Oxygen Permeability:

VALUE METHOD

21.4 x 10 11 (cm²/sec) Fatt (boundary corrected, edge corrected) (ml O<sub>2</sub>/ml x mm Hg) at 35°C

28.0 x 10 <sup>11</sup> (cm²/sec) Fatt (boundary corrected, non-edge corrected) (ml O₂/ml x mm Hg) at 35°C

#### **AVAILABLE LENS PARAMETERS**

The 1-DAY ACUVUE® DEFINE™ Contact Lenses are hemispherical shells of the following dimensions:

Diameter: 14.20 mm

Center Thickness: Low minus lens-varies with power (e.g., -3.00D, 0.084 mm)

Plus lens-varies with power (e.g., +1.00D, 0.130 mm)

creams, deodorants or sprays in the eyes or on the lenses. It is best to put on lenses before putting on makeup. Water-based cosmetics are less likely to damage lenses than oil-based products.

- DO NOT touch contact lenses with the fingers or hands if the hands are not free of foreign
  materials, as microscopic scratches of the lenses may occur, causing distorted vision and/or
  injury to the eye.
- Carefully follow the handling, application, removal, cleaning, disinfecting, storing and wearing
  instructions in the "Patient Instruction Guide" for the 1-DAY ACUNUE® DEFINE™ Contact Lenses
  and those prescribed by the Eye Care Professional.
- · Always handle lenses carefully and avoid dropping them.
- Never use tweezers or other tools to remove lenses from the lens container unless specifically indicated for that use. Slide the lens up the side of the bowl until it is free of the container.
- · Do not touch the lens with fingernails.

#### Lens Wearing Precautions:

- Due to the reduction in light transmittance with cosmetically tinted lenses, some patients may experience visual symptoms while wearing the 1-DAY ACUVUE® DEFINE™ Contact Lenses. In addition, some patients may experience peripheral awareness due to the opaque iris pattern.
- If the lens sticks (stops moving) on the eye, follow the recommended directions in "Care for a Sticking (Non-Moving) Lens". The lens should move freely on the eye for the continued health of the eye. If non-movement of the lens continues, the patient should be instructed to immediately consult the Eye Care Professional.
- Never wear lenses beyond the period recommended by the Eye Care Professional.
- The patient should be advised to never allow anyone else to wear their lenses. They have been
  prescribed to fit their eyes and to correct their vision to the degree necessary. Sharing lenses
  greatly increases the chance of eye infections.
- If aerosol products, such as hair spray, are used while wearing lenses, exercise caution and keep eyes closed until the spray has settled.
- Avoid all harmful or irritating vapors and fumes while wearing lenses.

#### Lens Care Precaution

The patient should be informed that no cleaning or disinfection is needed when lenses are worn
for daily disposable wear. Patients should always dispose of lenses when removed and have
spare lenses or spectacles available.

#### Other Topics to Discuss with Patients:

- · Always contact the Eye Care Professional before using any medicine in the eyes.
- Certain medications, such as antihistamines, decongestants, diuretics, muscle relaxants, tranquilizers and those for motion sickness may cause dryness of the eye, increased lens awareness

Base Curve: 8.5 mm

Power Range: -9.00D to -6.50D (in 0.50D increments)

-6,00D to -0,25D (In 0.25D increments) 0.00 to +1,00D (In 0.50D increments)

#### TRANSMITTANCE CURVES

1-DAY ACUVUE® DEFINE™ Brand Contact Lenses with LACREC 24 yr. old human cornea and 25 yr. old human crystalline lens.



\*The data are representative measurements taken through the central 3-5 r thinnest marketed lens (-3.00D lens, 0.084 mm center thickness).

WARNING: UV absorbing contact lenses are NOT substitutive UV absorbing eyewear, such as UV absorbing goggles because they do not completely cover the eye and surroup patient should continue to use UV absorbing eyewear as o

<sup>1</sup> Lerman, S., Radient Energy and the Eye, MacMillan, New York, 1990, p. 58, figure 2-21

<sup>2</sup> Waxler, M., Hitchins, V.M., Optical Radiation and Visual Health, CRC Press, Boca Raton, Florida

or blurred vision. Should such conditions exist, proper remedial measures Depending on the severity, this could include the use of lubricating drops use with soft contact lenses or the temporary discontinuance of contact is medication is being used.

- Oral contraceptive users could develop visual changes or changes in lens contact lenses. Patients should be cautioned accordingly.
- As with any contact lens, follow-up visits are necessary to assure the con patient's eyes. The patient should be instructed as to a recommended follows.

### Who Should Know That the Patient is Wearing Contact Le

- Patients should inform all doctors (Health Care Professionals) about being
- Patients should always inform their employer of being a contact lens wea require use of eye protection equipment or may require that the patient n

#### ADVERSE REACTIONS

The patient should be informed that the following problems may wearing contact lenses:

- The eye may burn, sting and/or itch.
- There may be less comfort than when the lens was first placed on the eye
- There may be a feeling of something in the eye (foreign body, scratched a
- There may be the potential for some temporary impairment due to periph peripheral comeal ulcers or corneal eroston. There may be the potential if observations, such as local or generalized edema, corneal neovasculariza injection, tarsal abnormalities, iritis and conjunctivitis; some of which are in low amounts.
- There may be excessive watering, unusual eye secretions or redness of the
- Poor visual acuity, blurred vision, rainbows or halos around objects, photo also occur if the lenses are worn continuously or for too long a time.

The patient should be instructed to conduct a simple 3-part self-least once a day. They should ask themselves:

- How do the lenses feel on my eves?
- How do my eyes look?
- Have I noticed a change in my vision?

If the patient reports any problems, he or she should be instructe REMOVE THE LENS. If the problem or discomfort stops, the patithe lens and place a new fresh k


| APPENDIX D: |
|------------------------------------------------------------------------|
| Near Logmar Visual Acuity Measurement Procedure |
| Lens Fitting Characteristics |
| Subject Reported Ocular Symptoms/Problems |
| Determination Of Distance Spherocylindrical Refractions |
| Biomicroscopy Scale |
| Distance And Near Visual Acuity Evaluation |
| Distance Logmar Visual Acuity Measurement Procedure |
| Measuring Pupil Diameter With Neuroptics VIP-200 Variable Pupillometer |
| Visual Acuity Chart Luminance And Room Illumination Testing |
| Qcsf Contrast Sensitivity |

NEAR LOGMAR VISUAL ACUITY MEASUREMENT PROCEDURE







LENS FITTING CHARACTERISTICS














SUBJECT REPORTED OCULAR SYMPTOMS/PROBLEMS



DETERMINATION OF DISTANCE SPHEROCYLINDRICAL REFRACTIONS



















BIOMICROSCOPY SCALE
















DISTANCE AND NEAR VISUAL ACUITY EVALUATION






CR-6396, v 2.0

JJVC CONFIDENTIAL







DISTANCE LOGMAR VISUAL ACUITY MEASUREMENT PROCEDURE








MEASURING PUPIL DIAMETER WITH NEUROPTICS VIP-200 VARIABLE PUPILLOMETER










VISUAL ACUITY CHART LUMINANCE AND ROOM ILLUMINATION TESTING

















QCSF CONTRAST SENSITIVITY















APPENDIX E: WORK AID: AST qVA-Custom 100











Work Aid: AST qVA-Custom 100





















APPENDIX F: WAVEFRONT AND TOPOGRAPHY MEASUREMENT USING VISIONIX VX118

# WORK AID: WAVEFRONT AND TOPOGRAPHY MEASUREMENT USING VISIONIX VX118 INSTRUMENT




Work Aid: Wavefront and Topography Measurement using Visionix VX118 instrument




Work Aid: Wavefront and Topography Measurement using Visionix VX118 instrument







Work Aid: Wavefront and Topography Measurement using Visionix VX118 instrument




Work Aid: Wavefront and Topography Measurement using Visionix VX118 instrument




Work Aid: Wavefront and Topography Measurement using Visionix VX118 instrument







APPENDIX G: COSMETIC FIT AND HULA HOOP







APPENDIX H: VISUAL EXPERIENCE WORK AID



#### PROTOCOL COMPLIANCE INVESTIGATOR(S) SIGNATURE PAGE

Protocol Number and Title: CR-6396 Objective Vision Evaluation of Two Cosmetic Contact Lenses

Version and Date: 2.0 29 January 2020

I have read and understand the protocol specified above and agree on its content.

I agree to conduct this study according to ISO 14155,<sup>1</sup> GCP and ICH guidelines,<sup>2</sup> the Declaration of Helsinki,<sup>3</sup> United States (US) Code of Federal Regulations (CFR),<sup>4</sup> and the pertinent individual country laws/regulations and to comply with its obligations, subject to ethical and safety considerations. The Principal Investigator is responsible for ensuring that all clinical site personnel, including Sub-Investigators adhere to all ICH<sup>2</sup> regulations and GCP guidelines regarding clinical trials during and after study completion.

I will assure that no deviation from or changes to the protocol will take place without prior agreement from the Sponsor and documented approval from the Institutional Review Board (IRB), except where necessary to eliminate an immediate hazard(s) to the trial participants.

I am responsible for ensuring that all clinical site personnel including Sub-Investigators adhere to all ICH<sup>2</sup> regulations and GCP guidelines regarding clinical trials during and after study completion.

All clinical site personnel involved in the conduct of this study have completed Human Subjects Protection Training.

I agree to ensure that all clinical site personnel involved in the conduct of this study are informed about their obligations in meeting the above commitments.

I shall not disclose the information contained in this protocol or any results obtained from this study without written authorization.

| Principal Investigator: | | |
|-------------------------|------------------------------------------|------|
| S | Signature | Date |
| | Name and Professional Position (Printed) | |
| Institution/Site: | | |
| | Institution/Site Name | |
| | Institution/Site Address | |